# Clinical Study Protocol

ZRHR-PK-02-JP

**Study title:** A single-center, open-label, randomized, controlled, crossover

study to investigate the nicotine pharmacokinetic profile and safety of Tobacco Heating System 2.2 (THS 2.2) following single use in smoking, healthy subjects compared to

conventional cigarettes and nicotine gum

Short title Nicotine pharmacokinetic profile and safety of the Tobacco

Heating System 2.2 (THS 2.2)

**Product name:** Tobacco Heating System 2.2 (THS 2.2)

**Sponsor:** Philip Morris Products S.A.

Quai Jeanrenaud 5 2000 Neuchâtel Switzerland

**Version number:** Final 1.0

**Date:** 21 June 2013

Authors: , PhD, Manager Clinical Science

, PhD, Biostatistician

, MD, Medical Safety Officer

, Medical Writer

#### **Confidentiality Statement**

Philip Morris Products S.A. ZRHR-PK-02-JP

Clinical Study Protocol Final 1.0 / 21 June 2013 Confidential


#### **SYNOPSIS**

Sponsor:

Philip Morris Products S.A.

#### Study Title:

A single-center, open-label, randomized, controlled, crossover study to investigate the nicotine pharmacokinetic profile and safety of Tobacco Heating System 2.2 (THS 2.2) following single use in smoking, healthy subjects compared to conventional cigarettes and nicotine gum.

Name of Product:

Tobacco Heating System 2.2 (THS 2.2)

Study Number and Acronym:

ZRHR-PK-02-JP, no acronym

### Primary Objective:

• To evaluate the rate and the amount of nicotine absorbed (as assessed by maximum plasma concentration  $[C_{max}]$  and area under the concentration-time curve [AUC] from start of product use to time of last quantifiable concentration  $[AUC_{(0-last)}]$ ) from THS 2.2 relative to conventional cigarettes (CC), following single use of THS 2.2 and CC.

#### Secondary Objectives:

- To determine if C<sub>max</sub> and AUC<sub>(0-last)</sub> of plasma nicotine of the THS 2.2 are higher relative to nicotine replacement therapy gum (NRT gum) following single use of the THS 2.2 and NRT gum.
- To evaluate the difference on nicotine pharmacokinetic (PK) absorption parameters (AUC from start of product use extrapolated to time of last quantifiable concentration to infinity [AUC<sub>(0-∞)</sub>] and partial AUC, where t' is the subject-specific time of maximum nicotine concentration following single use of the CC or NRT gum [AUC<sub>(0-t')</sub>]) between the THS 2.2 and CC, as well as the THS 2.2 and NRT gum.
- To evaluate the time to the maximum concentration (t<sub>max</sub>) of plasma nicotine for the THS 2.2 as compared to CC and to determine if the t<sub>max</sub> for THS 2.2 is shorter as compared to NRT gum.
- To describe the terminal half-life  $(t_{1/2})$  of nicotine for the THS 2.2, CC, and NRT gum.
- To describe the differences on urge-to-smoke over time between the THS 2.2 and CC, as

Philip Morris Products S.A.

Clinical Study Protocol Final 1.0 / 21 June 2013 

ZRHR-PK-02-JP

well as between the THS 2.2 and NRT gum.

- To describe product evaluation in the THS 2.2 and CC users.
- To describe the levels of carbon monoxide (CO) exposure for the THS 2.2, as compared to CC and NRT gum users.
- To monitor the safety during the study.

### **Primary Endpoints**:

- Primary nicotine PK parameters (THS 2.2 vs. CC):
  - o C<sub>max</sub>.
  - o AUC<sub>(0-last)</sub>.

Evaluation criterion: The study will be considered successful if the 95% confidence intervals (CI) of the THS 2.2:CC ratio for the primary nicotine PK parameters are estimated with a precision of  $\pm 20\%$ .

### Secondary Endpoints:

- Primary nicotine PK parameters (THS 2.2 vs. NRT gum)
- Secondary nicotine PK parameters:
  - $\circ$  AUC<sub>(0- $\infty$ )</sub>.
  - o Partial AUC<sub>(0-t')</sub>.
  - $\circ$   $t_{\text{max}}$ .
  - o  $t_{1/2}$ .
  - Subjective smoking effects:
    - Urge-to-smoke questionnaire (Questionnaire of Smoking Urges brief [QSU-brief]).
    - Product evaluation questionnaire (Modified Cigarette Evaluation Questionnaire [MCEQ]).
  - CO exposure biomarkers: levels of exhaled CO and carboxyhemoglobin (COHb) in blood.
  - Safety variables:
    - o Incidence of adverse events (AEs)/serious adverse events (SAEs), and including THS 2.2 malfunction/misuse.
    - o Respiratory symptoms: cough assessment by visual analogue and Likert scales and one open question.


- Vital signs.
- o Spirometry.
- o Electrocardiogram (ECG).
- o Clinical chemistry, hematology, and urine analysis safety panel.
- o Physical examination.
- Concomitant medications

#### Additional Study Assessments:

- Serology for human immunodeficiency virus 1/2 and Hepatitis B and C.
- Urine pregnancy test (females only), urine cotinine test, urine drug screen.
- Alcohol breath test.
- Chest X-ray.
- Nicotine dependence to be assessed with the Fagerström Test for Nicotine Dependence revised version.
- Cytochrome P450 2A6 (CYP2A6) activity (nicotine metabolic molar ratio) in plasma.

### Study Design:

This is a randomized, controlled, 2-period, 4-sequence, single-use crossover study. An incomplete block design is adopted, where each subject will receive only two of the three products (Figure S1):

- THS 2.2.
- CC.
- NRT gum.

ZRHR-PK-02-JP

Figure S1: Study Design

- Cross over with incomplete block design, 4 sequences
- · 62 smokers to be randomized



Abbreviations: THS: Tobacco Heating System; CC = conventional cigarette; NRT = Nicotine Replacement Therapy

A Screening Visit will be conducted within 4 weeks prior to Admission to the investigational site (Day -29 to Day -2) (Figure S1). A demonstration of the THS 2.2 product and the NRT gum will also be done by the site study collaborator during the Screening Visit. Subjects will be admitted to the clinic on Day -1. On Day -1, as the last procedure of the eligibility assessments on that day, all subjects will undergo a product test prior to enrolment, first THS 2.2 (using of up to 3 Tobacco Sticks) and subsequently NRT gum. In female subjects, the urine pregnancy test must be negative before any product test is performed with either the THS 2.2 or the NRT gum. After all inclusion and exclusion criteria have been satisfactorily met, only subjects willing and ready to use both the THS 2.2 and the NRT gum products can be enrolled. Screening procedures do not necessarily have to be conducted on the same day.

The confinement period will then consist of 2 periods (Period 1, Period 2) with each period consisting of at least 24-hour nicotine wash-out (nicotine abstinence) and 1 day of single product use.

Period 1: Day 0: Wash-out; Day 1: single product use (THS 2.2 /CC/NRT gum).

<u>Period 2:</u> Day 2: Wash-out; Day 3: single product use (THS 2.2 /CC/NRT gum).

| Philip Morris Products S.A. | Clinical Study Protocol | Confidential |
|-----------------------------|--------------------------|---------------|
| ZRHR-PK-02-JP | Final 1.0 / 21 June 2013 | |

In total, 62 eligible, healthy smoking subjects will be randomized into one of the 4 sequences:

```
Sequence 1: THS 2.2 \rightarrow CC (N=22)

Sequence 2: CC \rightarrow THS 2.2 (N=22)

Sequence 3: THS 2.2 \rightarrow NRT gum (N=9)

Sequence 4: NRT gum \rightarrow THS 2.2 (N=9)
```

Subjects will be discharged (time of discharge) from the investigational site in the morning of Day 4 after performance of the Day of Discharge assessments.

<u>From the time of discharge until Day 11</u>: A 7-day safety follow-up will be done for the recording of spontaneously reported new AEs and SAEs, and the active follow-up of ongoing AEs/SAEs by the site.

### Study Population and Main Criteria for Inclusion:

A total of 62 smoking, but healthy adult Japanese subjects, meeting the following main inclusion criteria:

- Subject is aged from 23 to 65 years (inclusive).
- Smoking, healthy subject as judged by the Investigator.
- Subject is Japanese.
- Subject smokes at least 10 commercially available CC per day (no brand restrictions) for the last 4 weeks, based on self-reporting.
- Subject does not plan to quit smoking in the next 3 months.
- Subject is ready to accept interruptions of smoking for up to 4 days.
- Subject is ready to accept using the THS 2.2 and the NRT gum product.

Each sex and each of the smoking strata (International Organization for Standardization [ISO] nicotine levels  $\leq$ 0.6 mg and 0.6 to 1 mg) will have a quota applied to ensure they represent at least 40% of the total study population. This will be applied to subjects randomized to sequence 1 and 2 and independently to subjects randomized to sequence 3 and 4. Subjects who do not complete the study after randomization will not be replaced.

### <u>Investigational Product, Dose, and Mode of Use:</u>

- Test Product: THS 2.2
- Reference Product, Dose, and Mode of Use:

Subject's own supply of commercially available preferred single brand CC

Philip Morris Products S.A. ZRHR-PK-02-JP

Clinical Study Protocol Final 1.0 / 21 June 2013 Confidential


### Reference Point Product (non-investigational):

Nicotine replacement therapy gum 2 mg Nicorette<sup>®</sup> chewed for  $35 \pm 5$  minutes. This will be supplied by the site and reimbursed by the Sponsor or designated Clinical Research Organization (CRO).

#### Duration of Study:

The entire study will last 14 to 41 days, including a Screening period of up to 4 weeks prior to Admission (Day -29 to Day -2), 6 days of confinement (Day -1 to time of discharge on Day 4), and 7 days of safety follow-up (from time of discharge until Day 11).

### Expected Duration of the Entire Study:

From 1<sup>st</sup> of July 2013 to 30<sup>th</sup> November 2013.

#### **Statistical Methods:**

All primary and secondary endpoints will be summarized with descriptive statistics. In addition, PK, subjective effects of smoking, and safety variables will be analyzed as follows.

Pharmacokinetics: the analysis populations for the PK endpoints will be composed of two analysis sets to allow the comparison between THS 2.2 and NRT gum separately from the comparison between THS 2.2 and CC. Only subjects without major protocol deviations will be included in the PK analysis sets.

Nicotine PK parameters will be derived from plasma nicotine versus time data using a non-compartmental technique.

An analysis of variance (ANOVA) will be conducted on logarithmically transformed  $AUC_{(0\text{-last})}$  and  $C_{max}$  primary endpoints. The model will include terms for sequence, subjects within sequence, period, and exposure group as fixed effect factors. The results of this analysis for each of  $AUC_{(0\text{-last})}$  and  $C_{max}$  will be presented in terms of adjusted geometric least square means and 95% CIs for the THS 2.2 :CC and THS 2.2:NRT gum ratios. The lower bound of the 95% CI of the THS 2.2:NRT gum ratio for  $C_{max}$  and  $AUC_{(0\text{-last})}$  will be compared with 1.00, to determine if the rate and the amount of nicotine absorbed of the THS 2.2 are higher relative to NRT gum

The  $AUC_{(0-\infty)}$ ,  $AUC_{(0-t')}$ , and  $t_{1/2}$  will be analyzed using the same approach adopted for the primary endpoints. The one-sided Wilcoxon Signed-Rank Test ( $\alpha$ =0.025) will be used to test if the  $t_{max}$  in THS 2.2 is shorter than in NRT gum. The median  $t_{max}$  differences between THS 2.2 and CC, as well as between THS 2.2 and NRT gum will be presented together with Hodges-Lehmann estimates of the 95% CI.

Subjective effects of smoking: mixed effects ANOVA using period, sequence, and product exposure as fixed effects and subjects within sequence as random effects will be adopted to analyze the domain scores of the product evaluation (MCEQ) questionnaire, for the comparison between THS 2.2 and CC. The same model will be evaluated for the analysis of

Clinical Study Protocol


ZRHR-PK-02-JP

Final 1.0 / 21 June 2013


urge-to-smoke (QSU-brief), including the assessment time points as repeated measurements. The results will be presented in terms of least square means and 95% CI for the THS 2.2 -CC and THS 2.2 -NRT gum differences.

<u>Safety:</u> The safety population will comprise all subjects who are exposed to THS 2.2 during the study, including the THS 2.2 test at admission.

Adverse event data will serve as the primary assessment of safety. All safety data will be listed and tabulated by sequence and by product use.

### Sample Size:

A total of 62 subjects will be randomized. This sample size is the sum of the sample size requirements for the THS 2.2:CC comparison and the THS 2.2:NRT gum comparison (as described in detail below).

The anticipated within-subject coefficients of variation for nicotine  $C_{max}$  and  $AUC_{(0-last)}$  are 36% and 21%, respectively.

The sample sizes of this study assume a drop-out rate no larger than 10%.

#### THS 2.2 :CC comparison

A total of 44 subjects are needed to estimate the mean  $C_{max}$  parameter ratio between THS 2.2 and CC with a 90% probability of obtaining a margin of error (95% CI) of at most  $\pm 20\%$ , assuming that THS 2.2 have a nicotine  $C_{max}$  similar to CC (ratio equal to 1.00). This sample size is sufficient to provide 90% probability of obtaining a margin of error of at most  $\pm 20\%$  for the AUC<sub>(0-last)</sub> ratio between THS 2.2 and CC, assuming a similar extent of nicotine absorption for the 2 products (ratio equal to 1.00).

#### THS 2.2 :NRT gum comparison

A total of 18 subjects are needed to estimate the mean  $AUC_{(0\text{-last})}$  parameter ratio between THS 2.2 and NRT gum with a precision allowing for the lower bound of the 95% CI exceeding 1.00, with 90% power, assuming a geometrical ratio between THS 2.2 and NRT gum of 1.28. This sample size is sufficient to provide 90% power of obtaining a lower bound of the 95% CI of  $C_{max}$  ratio between THS 2.2 and NRT gum, exceeding 1.00, assuming a geometrical mean ratio between THS 2.2 and NRT gum of 2.00.

### **TABLE OF CONTENTS**

| SY | NOPS | SIS | 2 |
|----|-------|-------------------------------------------------------|----|
| T | ABLE | OF CONTENTS | 9 |
| LI | ST OF | ABBREVIATIONS AND DEFINITIONS OF TERMS | 13 |
| 1 | ETI | HICS AND REGULATIONS | 19 |
| | 1.1 | Institutional Review Board Approval | 19 |
| | 1.2 | Ethical Conduct of the Study | 20 |
| | 1.3 | Subject Information and Consent | 20 |
| | 1.4 | Good Clinical Practice and Regulatory Requirements | 21 |
| 2 | INT | RODUCTION | 22 |
| | 2.1 | Background | 22 |
| | 2.2 | Purpose of the Study | 24 |
| | 2.3 | Anticipated Benefits and Risks | 24 |
| 3 | STU | JDY OBJECTIVES | 26 |
| | 3.1 | Primary Objective | 26 |
| | 3.2 | Secondary Objectives | 26 |
| | 3.3 | Primary Endpoints | 27 |
| | 3.4 | Secondary Endpoints | 27 |
| | 3.5 | Exploratory Endpoints | 28 |
| 4 | INV | ESTIGATIONAL PLAN | 29 |
| | 4.1 | Overall Study Design and Plan | 29 |
| | 4.2 | Rationale for Study Design and Control Group(s) | 32 |
| | 4.3 | Study Duration | 32 |
| | 4.4 | Appropriateness of Measurement | 33 |
| 5 | STU | JDY POPULATION | 34 |
| | 5.1 | Selection of Study Population | 34 |
| 6 | INV | ESTIGATIONAL PRODUCTS AND REFERENCE POINT PRODUCT | 41 |
| | 6.1 | Description | 41 |
| | 6.2 | Use of Investigational and Reference Point Products | 44 |
| | 6.3 | Method for Assigning Subjects to Study Arms | 46 |
| | 6.4 | Blinding | 46 |
| | 6.5 | Investigational Product Accountability and Compliance | 47 |
| | 6.6 | Restrictions | 48 |

ZRHR-PK-02-JP

Final 1.0 / 21 June 2013


| 7 | STU | DY PROCEDURES | 52 |
|---|---|---|---|
| | 7.1 | Informed Consent. | 52 |
| | 7.2 | Smoking Cessation Advice and Debriefing | 52 |
| | 7.3 | Support during Smoking Abstinence/Periods of Reduced Smoking | 53 |
| | 7.4 | Clinical Assessments | 53 |
| | 7.5 | Biomarker Assessment. | 56 |
| | 7.6 | Laboratory Assessments | 58 |
| | 7.7 | Sample Handling, Storage, and Shipment | 60 |
| | 7.8 | Questionnaires | 61 |
| 8 | ADV | /ERSE EVENTS | 64 |
| | 8.1 | Definitions | 64 |
| | 8.2 | Assessment of Adverse Events | 65 |
| | 8.3 | Reporting of Serious Adverse Events | 67 |
| | 8.4 | Reporting of Other Events Critical to Safety Evaluations | 68 |
| | 8.5 | Actions and Follow-up. | 70 |
| 9 | STU | DY ACTIVITIES | 72 |
| | 9.1 | Screening Visit | 72 |
| | 9.2 | Admission | 73 |
| | 9.3 | Investigational Period | 75 |
| | 9.4 | Day of Discharge | 81 |
| | 9.5 | Safety Follow-up Period | 83 |
| | 9.6 | Early Termination Procedures | 83 |
| 10 | QUA | ALITY CONTROL AND QUALITY ASSURANCE | 84 |
| | 10.1 | Monitoring | 84 |
| | 10.2 | Training of Study Collaborator | 85 |
| | 10.3 | Audits and Inspections | 85 |
| 11 | DAT | TA MANAGEMENT ACTIVITIES | 86 |
| | 11.1 | Data Capture | 86 |
| | 11.2 | Data Handling | 87 |
| 12 | PLA | NNED STATISTICAL METHODS | 89 |
| | 12.1 | General Considerations | 89 |
| | 12.2 | Determination of Sample Size and Power Consideration | |
| | 12.3 | Analysis Populations | 91 |
| | 12.4 | Demographics and Baseline Characteristics | 92 |

| Philip Morris P | roducts S.A. Clinical Study Protocol | Confidential |
|---|---|---|
| ZRHR-PK-02-J | P Final 1.0 / 21 June 2013 | |
| 12.5 P | rimary Endpoints | 92 |
| 12.6 S | econdary Endpoints | 93 |
| 12.7 E | xploratory Analyses | 96 |
| 12.8 In | nterim Analysis | 96 |
| 13 ADMIN | NISTRATIVE CONSIDERATIONS | 96 |
| 13.1 P | rincipal Investigators and Study Administrative Structure | 96 |
| (b) (4) | | 98 |
| 13.2 S | ubject Confidentiality | 98 |
| 13.3 A | access to Source Documentation | 99 |
| 13.4 R | ecord Retention | 99 |
| 13.5 C | Clinical Study Report | 101 |
| 13.6 F | inancial Disclosure | 101 |
| 13.7 P | ublication and Disclosure Policy | 101 |
| 13.8 In | nsurance | 102 |
| 14 REFER | ENCE LIST | 103 |


#### LIST OF IN-TEXT TABLES AND FIGURES

| Table 1 | Measured aerosol fractions for the THS Tobacco Sticks | 42 |
|---|---|---|
| Table 2 | Drugs and Substances Considered Interacting with CYP2A6 | 50 |
| Table 3. | Clinical Laboratory Parameters for Safety Panel | 59 |
| Table 4 | Time Schedule – Screening Visit | 72 |
| Table 5. | Time Schedule – Day -1 Admission | 74 |
| Table 6. | Time Schedule – Day 0 Washout. | 75 |
| Table 7. | Time Schedule – Day 2 Washout. | 77 |
| Table 8. | Time Schedule – Day 1 and Day 3 Product Use | 79 |
| Table 9. | Time Schedule – Day 4 Discharge | 82 |
| Figure 1. | Study Flow Chart | 31 |
| LIST OF APPEN | NDICES | |
| Appendix 1 | Schedule of Events | 109 |
| Appendix 2 | Participating Laboratories | 113 |
| Appendix 3 | Investigational Product and Instructions for Use | 114 |
| Appendix 4 | THS Package Label | 115 |
| Appendix 5 | Abnormal Laboratory Values | 118 |

Philip Morris Products S.A.

Clinical Study Protocol


ZRHR-PK-02-JP

Final 1.0 / 21 June 2013


### LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

#### **Abbreviations**

ADL Activities of daily living

AE Adverse event

ALT Alanine aminotransferase

ANOVA Analysis of variance

AST Aspartate aminotransferase

AUC Area under the concentration-time curve

 $AUC_{(0-\infty)}$  Area under the concentration-time curve from start of product use extrapolated

to time of last quantifiable concentration to infinity

AUC<sub>(0-last)</sub> Area under the concentration-time curve from start of product use to time of

last quantifiable concentration

AUC<sub>(0-t')</sub> Partial AUC, where t' is the subject-specific time of maximum nicotine

concentration following single use of conventional cigarettes or NRT gum

BMI Body mass index

CC Conventional cigarette(s)

CD Compact disc

CI Confidence Interval

C<sub>last</sub> Last quantifiable concentration

C<sub>max</sub> Maximum plasma concentration

CO Carbon monoxide

Philip Morris Products S.A. Clinical Study Protocol Confidential ZRHR-PK-02-JP Final 1.0 / 21 June 2013 

COHb Carboxyhemoglobin

CRA Clinical Research Associate

CRO Contract Research Organization

CSR Clinical Study Report

CTCAE Common Terminology Criteria for Adverse Events and Common Toxicity

Criteria

CTMS Clinical Trial Management System

CV Coefficient of variation

CYP2A6 Cytochrome P450 2A6

DMP Data Management Plan

ECG Electrocardiogram

eCRF Electronic Case Report Form

EOS End of Study (referring to each subject's individual last study visit)

ePRO Electronic patient reported outcome

FDA Food and Drug Administration

 $FEV_1$  Forced expiratory volume in 1 second

FTND Fagerström Test for Nicotine Dependence

FVC Forced vital capacity

GCP Good Clinical Practice

HIV Human immunodeficiency virus

Philip Morris Products S.A.

Clinical Study Protocol


ZRHR-PK-02-JP

Final 1.0 / 21 June 2013


HPHC Harmful and potentially harmful constituents

IB Investigator's Brochure

ICF Informed consent form

ICH International Conference on Harmonization

IP Investigational Product

IRB Institutional Review Board

ISO International Organization for Standardization

IV Intravenous

LLN Lower limit of the normal range

LLOQ Lower limit of quantification

MCEQ Modified Cigarette Evaluation Questionnaire

MedDRA Medical Dictionary for Regulatory Activities

MRTP Modified risk tobacco product

n Number of subjects

NRT gum Nicotine replacement therapy gum

PK Pharmacokinetic(s)

PMI Philip Morris International

QC Quality control

QSU-brief Questionnaire of Smoking Urges brief

SA Smoking abstinence

SAE Serious adverse event

Philip Morris Products S.A.

ZRHR-PK-02-JP

Clinical Study Protocol Final 1.0 / 21 June 2013 Confidential


SAP Statistical Analysis Plan

SHM Sample handling manual

SOP Standard Operating Procedure

T Time point

 $T_0$  Time point of first product use during study day

t<sub>1/2</sub> Terminal half-life

THS 2.2 Tobacco Heating System 2.2

t<sub>max</sub> Time to the maximum concentration

ULN Upper limit of the normal range

ULOQ Upper limit of quantification

VAS Visual Analogue Scale

WBC White blood cell (count)

WHO World Health Organization

 $\lambda_z$  Terminal elimination rate constant

### **Explanations of Terms**

The following special terms are used in this protocol:

CC The term 'conventional cigarette' refers to manufactured and

commercially available cigarettes and excludes hand-rolled cigarettes, cigars, pipes, bidis, and other nicotine-containing

products. Conventional cigarettes are designated "CC".

Charger: The function of the Charger (Model 4) is to recharge the Holder

after use. It contains a battery with sufficient capacity to recharge the Holder approximately 20 times. It is a convenient size to carry around, and can itself be recharged from a mains power source.

Day of Discharge Day 4.

End of Study End of Study is defined as the last day of the 7-day safety

follow-up subsequent to discharge from the clinic.

Enrolment On Day -1 for eligible subjects after all applicable inclusion and

exclusion criteria have been satisfactorily met and the subject is willing and ready to use both the Tobacco Heating System 2.2 THS 2.2 and nicotine replacement therapy gum (NRT gum). The test of both THS 2.2 and NRT gum are the last assessments prior to

enrolment.

Investigator Principal Investigator or sub-Investigator

First product use time Start of produ

point

Start of product use for THS 2.2 is defined as the time of the first puff. The start time for CC corresponds to the lighting of the CC, and the start time of the NRT gum product is the time of NRT gum

intake.

Randomization Assignment to product on Day 0 utilizing an Interactive Web and

Voice Response System.

Safety follow-up After the time of discharge, a 7-day safety follow-up will be done

for the recording of spontaneously reported new adverse events (AEs)/serious adverse events (SAEs) and the active follow-up of ongoing AEs/SAEs by the site. In general any AE will be followed up until resolved, stabilized i.e., no worsening of the event or a

plausible explanation for the event has been found.

| Philip Morris Products S.A. | Clinical Study Protocol | Confidential |
|---|---|---|
| ZRHR-PK-02-JP | Final 1.0 / 21 June 2013 | |
| Screening failure | Subjects who do not meet the entry criteria fr form (ICF) signature to the time of enrolment screening failure and will be replaced by other | will be considered a |
| THS Tobacco Stick<br>Holder (Holder) | The function of the Holder (Model 4.2) is Stick, delivering an aerosol to the user. The powered from an internal battery which delive minutes (allowing complete use of a single To | e electrical heating is ers power for about 6 |
| THS Tobacco Stick | The Tobacco Stick (product code C3) cont when heated, generates an aerosol. It is custon with the Holder. | · |

Clinical Study Protocol Final 1.0 / 21 June 2013


#### 1 ETHICS AND REGULATIONS

### 1.1 Institutional Review Board Approval

Prior to the start of the study, the clinical study protocol, together with its associated documents (informed consent form [ICF] which includes both subject information sheet and informed consent, subject recruitment procedures [e.g., advertisements], written information to be provided to the subjects, Investigator's Brochure [IB], available safety information, the Principal Investigator's curriculum vitae and/or other evidence of qualifications, the list of sub-Investigators and any other documents requested by the Institutional Review Board [IRB]), will be submitted for review and approval to the relevant IRB. The IRB shall be appropriately constituted and perform its functions in accordance with the International Conference on Harmonisation (ICH) Tripartite Guidance for Good Clinical Practice (GCP), Ministerial Ordinance on GCP for Drugs, and local requirements, as applicable.

In accordance with GCP, a written confirmation of the IRB approval should be provided to the Sponsor. This should identify the study (Principal Investigator's name, study number, and title) and the documents that have been approved by the IRB, with dates and version numbers, as well as the date of approval. The composition of the IRB, including the name and occupation of the chairperson, should be supplied to the Sponsor together with a GCP compliance statement.

The written approval from the IRB will be filed in the Investigator file, and another original copy will be filed in the Study Master File at the Sponsor or designated organization. The study must not start before the Sponsor has obtained written confirmation of favorable opinion/approval from the concerned IRB.

Any substantial change or addition to this protocol will require a written protocol amendment that must be approved by the Sponsor and the Principal Investigator. All amendments will be submitted to the IRB, and substantial amendments will only be implemented after approval by the IRB.

These requirements for approval should in no way prevent any action from being taken by the Principal Investigator or sub-Investigator (Investigator) or by the Sponsor in order to eliminate immediate hazards to the subjects. If such a change to the protocol is felt to be necessary by the Investigator, and is implemented for safety reasons, the Sponsor and the IRB should be informed immediately.

Relevant safety information will be submitted to the IRB during the course of the study in accordance with national regulations and requirements.

Clinical Study Protocol Final 1.0 / 21 June 2013


# 1.2 Ethical Conduct of the Study

The study will be performed in accordance with ethical principles that have their origin in the Declaration of Helsinki, 2008 and are consistent with ICH/GCP, Ethical Guidelines for Clinical Studies (Ministry of Health, Labour and Welfare, 2003 [as last amended on July 31, 2008]), Ministerial Ordinance on Good Clinical practice for Drugs (Ministry of Health, Labour and Welfare, 1997 (as last amended by the Ordinance of Ministry of Health, Labour and Welfare No. 161 of December 28, 2012)), and applicable regulatory principles.

The Principal Investigator agrees to conduct the clinical study in compliance with the protocol agreed upon with the Sponsor and approved by the IRB. The Principal Investigator and the Sponsor must sign the protocol (and protocol amendments, if applicable) to confirm this agreement. A copy of the Declaration of Helsinki, 2008 should be located in the Investigator's Study File.

### 1.3 Subject Information and Consent

### 1.3.1 Study Consent/Subject Information Sheet

Before or at the Screening Visit, the Investigator will ensure each subject is given full and adequate oral and written information about the nature, purpose, possible risks and benefits of the study, and the Investigator will answer all questions the subject might have to his/her full satisfaction. The subject will have sufficient time for consideration of his/her participation in the study and will be notified that he/she is free to discontinue his/her participation at any time. Once the subject has received all necessary information, and if he/she agrees to participate, this will be documented in the ICF by the date and signature of both the subject and the person who conducted the informed consent discussion. No study-specific procedures will be performed before the ICF has been signed.

The original, dated and signed ICF(s) must be kept in the Investigator file at the site, and a copy must be given to the subject.

The subject will be informed that additional data analyses not mentioned in the protocol or the statistical analysis plan might be performed with the collected data at a later time. If any additional analyses will be performed, they will fully be covered by data confidentiality, as for the main analyses described in this protocol.

### 1.3.2 Amendment to the Informed Consent Form/Subject Information Sheet

If a protocol amendment is required, or if new information regarding the risk profile of the Investigational Product (IP) becomes available, an amendment may be required to the ICF. If revision of the ICF is necessary, the Principal Investigator will, with the support of the

Philip Morris Products S.A. ZRHR-PK-02-JP

Clinical Study Protocol Final 1.0 / 21 June 2013 Confidential


Sponsor, ensure that the documents have been reviewed and approved by a relevant IRB before subjects are required to re-sign the ICF.

### 1.4 Good Clinical Practice and Regulatory Requirements

The procedures set out in this clinical study protocol pertaining to the conduct, evaluation, and documentation of this study are designed to ensure that the Sponsor, its authorized representative, and the Principal Investigator abide by the principles of the ICH guidelines on GCP. These guidelines apply specifically to pharmaceutical development, but nevertheless provide a robust and ethical framework for conducting clinical studies of tobacco products. In addition, the Investigator will carry out the clinical study in accordance with GCP and Ethical Guidelines for Clinical Studies.

Clinical Study Protocol Final 1.0 / 21 June 2013 Confidential


#### 2 INTRODUCTION

### 2.1 Background

### 2.1.1 Smoking-Related Diseases and Harm Reduction Strategy

Cigarette smoking causes pulmonary and cardiovascular diseases and other serious diseases in smokers (U.S. Department of Health and Human Services, 2010). The effects of smoking and smoking cessation on mortality from cardiovascular disease among the Japanese population were investigated in cohort studies in Japan. These studies confirmed the association between smoking and mortality from cardiovascular disease and highlighted the importance of smoking cessation at any age to prevent cardiovascular disease in the Japanese population (Honjo et al., 2010a, Iso et al., 2005). In 2000 in Japan, the proportion of adult deaths due to smoking ranges from 20.0% to 24.9% in males and from 10.0% to 14.6% in females. In 2007, Japan became part of the top 5 conventional cigarette (CC)-consuming countries with a consumption of 234 billion annually in 2009 (World Lung Foundation, 2012). There is no safe cigarette and the best way for smokers to reduce the adverse health consequences of smoking is to quit. Despite the risks which are attributable to smoking, some smokers cannot refrain from smoking or decide to continue smoking. To those smokers who are not able or not willing to quit, Philip Morris International (PMI) is developing alternative approaches by developing products with the potential to reduce the risks of tobacco-related diseases. These products are now referred to by the US Food and Drug Administration (FDA) as modified risk tobacco products (MRTPs) (FDA, 2012c).

The challenge in developing and commercializing MRTPs is two-fold, i.e. developing tobacco products that are shown to reduce risk and that are acceptable to smokers as substitutes for CCs. PMI is developing candidate MRTP that provide an inhalation experience without combustion. The novel approach to achieve this is by heating tobacco at significantly lower temperatures than required for CC.

PMI's approach to scientifically assessing the risk-reduction potential of its candidate MRTPs is described in the reference document (PMI White Paper Docket). Smoking cessation is the only intervention proven to reduce the risk of smoking-related diseases in smokers. Accordingly, PMI utilizes smoking cessation/smoking abstinence (SA) as the benchmark for assessing the risk reduction potential of its candidate MRTPs. The Institute of Medicine observed that cessation is the "gold standard" for assessing risk reduction, and that "the closer risks and exposures from the MRTP are to cessation products, the more confident a regulator can be of achieving a net public health benefit" (Institute of Medicine, 2012). PMI has already conducted studies and plans to conduct further clinical studies which observe measurable changes in blood chemistry, risk factors and health effects in smokers


who switch to a candidate MRTP, comparing the changes with those observed in both smokers who continue smoking CC and smokers who stop using tobacco products. Longer-term data from adults who continue to use the candidate MRTP can further substantiate reductions in individual risk in smokers and population harm.

### 2.1.2 Description of the Product and Scientific Findings

Thousands of chemicals - "smoke constituents" - are formed when tobacco is burned or combusted. More than 5,300 smoke constituents have been identified (Rodgman and Perfetti, 2009), and more than 100 of them have been categorized as harmful and potentially harmful constituents (HPHC) (FDA, 2011). There is no convincing evidence that selective reduction of smoke constituents can reduce tobacco related diseases (Hatsukami et al., 2007). Philip Morris International's focus has been the development of products that do not combust tobacco but which replicate the "smoking experience" traditionally obtained with CC, as much as possible. Our approach limits pyrolysis and combustion, by heating tobacco at significantly lower temperatures than CC. Philip Morris International believes that such products present the best opportunity for reducing harm because they produce vastly lower levels of harmful smoke constituents and are more likely to be accepted by smokers as substitutes for CCs. Important to this effort has been providing nicotine in a way that closely parallels CC.

The product developed by PMI, and to be assessed in this study, is the Tobacco Heating System 2.2 (THS 2.2). With this product, the heating of the tobacco is maintained below 400°C, a temperature much lower than what is observed for CC, which can reach 900°C. The THS 2.2 is composed of the 'THS Tobacco Stick Holder', dedicated special Tobacco Sticks made of conventional tobacco, a Charger, and different accessories. The energy of the THS Tobacco Stick Holder is sufficient to maintain approximately a 6 minute session. Unlike CC, the Tobacco Sticks do not burn down during their consumption and their lengths remain constant after use.

The non-clinical assessment of THS 2.2 and its predecessors including THS 1.0 described in the Investigator's Brochure (PMI, 2013b) supports the initiation of the clinical studies. No new or increased toxicological hazard in the product's aerosol was detected, compared with CC smoke. The aerosol was chemically analyzed confirming that none of the determined HPHCs in the THS 2.2 were increased compared to the CC. The biological activity was tested in a number of *in vitro* assays to assess the cytotoxicity and the genotoxicity of the aerosol fractions total particulate matter (TPM) and gas vapor phase (GVP). *In vitro* and *in vivo* results corroborated the concept that absence of combustion when consuming tobacco substantially lowers toxic effects seen in these biological models. Further details are given in the Investigator's' Brochure (PMI, 2013b).


Several clinical studies have been conducted on THS 1.0, an earlier development version of THS 2.2, in Europe, Asia, Africa and the United States. All studies showed reductions in exposure to the majority of measured HPHCs from both aerosol fractions, TPM and GVP, in subjects who used the THS 1.0 as compared to subjects continuing smoking CC, both, in controlled and ambulatory conditions.

The previous version of THS 2.2, namely THS 2.1 was tested in two exploratory clinical studies to measure the nicotine plasma kinetic profile (PK) (www.clinicaltrials.gov identifier: NCT01780688) and to assess the reduction of exposure to HPHCs (www.clinicaltrials.gov identifier: NCT01780714) when switching from CC to THS 2.1. The observed nicotine plasma PK profile for THS 2.1 was similar to CC as well, there were significant reductions in the exposure to the majority of selected HPHCs. Clinical studies conducted so far revealed no safety concern for either of the previous version of THS 2.2 tested. Further details on the clinical data are provided in the Investigators' Brochure (PMI, 2013b.).

#### 2.2 **Purpose of the Study**

The purpose of this clinical study is to compare the profile of nicotine uptake (rate and extent of nicotine absorbed) after single use of switching from conventional cigarettes (CC) to THS 2.2 and CC in smoking Japanese healthy smokers. THS 2.2 will also be compared with the nicotine replacement therapy gum (NRT gum), used as a reference point.

#### 2.3 **Anticipated Benefits and Risks**

#### 2.3.1 **Anticipated Benefits**

In Japan, research conducted by the Ministry of Health, Labour and Welfare has shown that 35.9% of male and 43.6% of female respondents over 20 years of age expressed the wish to quit smoking (International Tobacco Online, 2012). In a large follow-up study of middle aged Japanese smokers, the predictors of smoking cessation were age, job, smoking habit, physical activity, health checkup participation, and health status (Honjo et al., 2010b). Advice on health risks associated with smoking and smoking cessation advice will be provided at Screening, at Admission, and at the Day of Discharge. The advice will follow the recommendations of the World Health Organization (WHO) (WHO, 2002) - "Evidence based Recommendations on the Treatment of Tobacco Dependence". Subjects who are motivated to quit smoking during the study will be given the opportunity to continue their smoking cessation attempt and will be referred to appropriate stop smoking services for continuing support and counseling at a higher level. Subjects who participate in this study will also benefit from repeated, detailed health check-ups, which may help to uncover undiagnosed medical conditions.


### 2.3.2 Anticipated Foreseeable Risks due to Study Procedures

- Risks related to blood sampling, e.g., excessive bleeding, fainting, hematoma, paresthesia, or infection.
- Risks related to chest X-rays, e.g., a small increase of risk to develop cancer later in life.
- Risks related to drug application as part of testing procedures (i.e. spirometry with short-acting bronchodilator at Screening) per study protocol and scientifically accepted standards.
- 2.3.3 Anticipated Foreseeable Risks due to Investigational Product (THS 2.2/CC) or Reference Point Product
- Change in smoking habits due to study requirements and related concomitant symptoms, (e.g., craving, withdrawal symptoms).

All risks related to study procedures, IP, or support for SA will be explained in detail to the subjects. Mitigation will include, but will not be limited to:

- Close monitoring and medical evaluation of potential safety signals throughout the study and follow-up.
- Using accepted research and scientific standards, (e.g., blood samples not to exceed local blood donation standards).
- Management and follow-up of adverse events (AEs)/serious adverse events (SAEs).
- Risks specific to the use of any NRT gum, as per the relevant summary of product characteristics.

#### 2.3.4 Unforeseeable Risks

As with any new IP, and the reference point product, there may be unforeseeable risks and hazards that could occur. The possibility of such will be explained at Screening and at Admission. Mitigation will include close monitoring and medical supervision to detect any unforeseeable risk or safety signals at the earliest possibility.


### 3 STUDY OBJECTIVES

### 3.1 Primary Objective

The primary objective of this study is:

• To evaluate the rate and the amount of nicotine absorbed (as assessed by maximum plasma concentration [C<sub>max</sub>] and area under the concentration-time curve [AUC] from start of product use to time of last quantifiable concentration [AUC<sub>(0-last)</sub>]) from THS 2.2 relative to CC, following single use of THS 2.2 and CC.

### 3.2 Secondary Objectives

The secondary objectives of this study are:

- To determine if  $C_{max}$  and  $AUC_{(0-last)}$  of plasma nicotine of the THS 2.2 are higher relative to NRT gum following single use of the THS 2.2 and NRT gum.
- To evaluate the difference on nicotine pharmacokinetic (PK) absorption parameters (AUC from start of product use extrapolated to time of last quantifiable concentration to infinity [AUC<sub>(0-∞)</sub>] and partial AUC, where t' is the subject-specific time of maximum nicotine concentration following single use of CC or NRT gum [AUC<sub>(0-t')</sub>] between the THS 2.2 and CC, as well as the THS 2.2 and NRT gum.
- To evaluate the time to the maximum concentration (t<sub>max</sub>) of plasma nicotine for the THS 2.2 as compared to CC and to determine if the t<sub>max</sub> for THS 2.2 is shorter as compared to NRT gum.
- To describe the terminal half-life  $(t_{1/2})$  of nicotine for the THS 2.2, CC, and NRT gum.
- To describe the differences on urge-to-smoke over time between the THS 2.2 and CC, as well as between the THS 2.2 and NRT gum.
- To describe product evaluation in the THS 2.2 and CC users.
- To describe the levels of carbon monoxide (CO) exposure for the THS 2.2, as compared to CC and NRT gum users.
- To monitor the safety during the study.


ZRHR-PK-02-JP

Final 1.0 / 21 June 2013


# 3.3 Primary Endpoints

- Primary nicotine PK parameters (THS 2.2 vs CC):
  - $\circ$   $C_{max}$
  - o AUC<sub>(0-last)</sub>.

#### Evaluation criterion:

The study will be considered successful if the 95% confidence intervals (CI) of the THS 2.2:CC ratio for the primary nicotine PK parameters are estimated with a precision of  $\pm 20\%$ .

### 3.4 Secondary Endpoints

- Primary nicotine PK parameters (THS 2.2 vs. NRT gum)
- Secondary nicotine PK parameters
  - $\circ$  AUC<sub>(0- $\infty$ ).</sub>
  - o Partial AUC<sub>(0-t')</sub>.
  - $\circ$   $t_{max}$
  - $\circ$   $t_{1/2}$
- Subjective smoking effects:
  - o Urge-to-smoke questionnaire (Questionnaire of Smoking Urges brief [QSU-brief]).
  - o Product evaluation questionnaire (Modified Cigarette Evaluation Questionnaire [MCEQ]).
- CO exposure biomarkers: levels of exhaled CO and carboxyhemoglobin (COHb) in blood.
- Safety variables:
  - o Incidence of AEs/SAEs and device events, including THS 2.2 malfunction/misuse.
  - o Respiratory symptoms: cough assessment by Visual Analogue Scale (VAS) and Likert scales and one open question.
  - o Vital signs.
  - o Spirometry.
  - o Electrocardiogram (ECG).
  - o Clinical chemistry, hematology, and urine analysis safety panel.
  - Physical examination.
  - Concomitant medications.

Philip Morris Products S.A. ZRHR-PK-02-JP

Clinical Study Protocol Final 1.0 / 21 June 2013 

### Additional Study Assessments:

- Serology for human immunodeficiency virus 1/2 and Hepatitis B and C.
- Urine pregnancy test (females only), urine cotinine test, urine drug screen.
- Alcohol breath test.
- Chest X-ray.
- Nicotine dependence to be assessed with the Fagerström Test for Nicotine Dependence (FTND) revised version.
- Cytochrome P450 2A6 (CYP2A6) activity (nicotine metabolic molar ratio) in plasma.

### 3.5 Exploratory Endpoints

There are no exploratory analyses planned.


4 INVESTIGATIONAL PLAN

### 4.1 Overall Study Design and Plan

This is a randomized, controlled, 2-period, 4-sequence, single use crossover study where each subject will receive two of the three products:

- THS 2.2.
- CC.
- NRT gum.

A Screening Visit will be conducted within 4 weeks prior to Admission to the investigational site (Day -29 to Day -2) (Figure 1). A demonstration of the THS 2.2 product and the NRT gum will also be done by the study site collaborator during the Screening Visit. Subjects will be admitted to the clinic on Day -1. On Day -1, as the last procedure of the eligibility assessments on that day, all subjects will undergo a product test prior to enrolment: first THS 2.2 and subsequently NRT gum (using up to 3 Tobacco Sticks). In female subjects, the urine pregnancy test must be negative before any product test is performed with either the THS 2.2 or the NRT gum. After all inclusion and exclusion criteria have been satisfactorily met, only subjects willing and ready to use both the THS 2.2 and the NRT gum products can be enrolled. Screening procedures do not necessarily have to be conducted on the same day.

The confinement period will then consist of 2 periods (Period 1, Period 2) with each period consisting of at least 24-hour nicotine wash-out (nicotine abstinence) and 1 day of single product use.

Period 1: Day 0: Wash-out; Day 1: single product use (THS 2.2 /CC/NRT gum).

Period 2: Day 2: Wash-out; Day 3: single product use (THS 2.2 /CC/NRT gum).

In total, 62 eligible, smoking subjects will be randomized into 1 of the 4 sequences:

Sequence 1: THS 2.2  $\rightarrow$  CC (N=22). Sequence 2: CC  $\rightarrow$  THS 2.2 (N=22). Sequence 3: THS 2.2  $\rightarrow$  NRT gum (N=9). Sequence 4: NRT gum  $\rightarrow$  THS 2.2 (N=9).

Philip Morris Products S.A.

Clinical Study Protocol


ZRHR-PK-02-JP

Final 1.0 / 21 June 2013


This procedure will lead to an incomplete block design with every subject being exposed to 2 of the 3 study products, as the comparison between NRT gum and CC will not be considered.

CC vs. THS 2.2 (N=22 in both sequence 1 and 2). (N=9 in both sequence 3 and 4). THS 2.2 vs. NRT gum

Each sex and each of the smoking strata (International Organization for Standardization [ISO] nicotine levels  $\leq 0.6$  mg and 0.6 to 1 mg) will have a quota applied to ensure they represent at least 40% of the total study population. This will be applied to subjects randomized to sequence 1 and 2 and independently to subjects randomized to sequence 3 and 4

Subjects will be discharged (time of discharge) from the investigational site in the morning of Day 4 after all examinations of the Day of Discharge have been conducted. After the time of discharge, a 7-day safety follow-up will be started for the recording of spontaneously reported new AEs/SAEs and the active follow-up of ongoing AEs/SAEs by the site. Any AE will, in general, be followed up until resolved, stabilized (i.e., no worsening of the event), or until a plausible explanation for the event has been found.


ZRHR-PK-02-JP

Figure 1. Study Flow Chart

- Cross over with incomplete block design, 4 sequences
- 62 smokers to be randomized



Abbreviations: THS: Tobacco Heating System; CC = conventional cigarette; NRT = Nicotine Replacement Therapy


### 4.2 Rationale for Study Design and Control Group(s)

The minimum age of 23 years age in the inclusion criteria was selected based on:

- The legal age of smoking in Japan is 20 years.
- To account for the 3 years of smoking history.

In this study, CCs (up to 1.0 mg nicotine ISO yield/CC) will be used as a reference product and a market-approved pharmaceutical NRT gum 2 mg (Nicorette<sup>®</sup>) will be used as non-investigational reference point. The NRT gum has been selected as the reference point, because of its availability over the market. The NRT gum will serve as a reference point for comparison with THS 2.2 for the following endpoints:

- Nicotine PK parameters.
- Urge-to-smoke.
- Safety profile.

The nicotine wash-out period was set to at least 24 hours (>5 x elimination  $t_{1/2}$ ) as the elimination  $t_{1/2}$  of nicotine in blood is around 2 hours in Caucasian smokers (Benowitz et al., 2009).

The use of estrogen contraceptive is known to accelerate nicotine clearance by 20% to 30% in women as compared to women who do not take such contraceptives (Benowitz et al., 2006). Therefore, for the purpose of this study, it is not allowed to use hormonal contraception containing estrogens. This also applies to hormone replacement therapy.

In this study, THS 2.2 will be tested against CC and NRT gum will be used as a reference point product.

Furthermore, CYP2A6 activity will be assessed in this study. Asians on average metabolize nicotine more slowly than Caucasians do, at least in part due to a high prevalence of the CYP2A6 alleles associated with reduced or absent enzyme activity (Matta et al., 2006).

# 4.3 Study Duration

The entire study per subject will last 14 to 40 days, including a Screening period of up to 4 weeks prior to Admission (Day -29 to Day -2), 6 days of confinement (Day -1 to morning of Day 4), and 7 days of safety follow-up (from time of discharge until Day 11). In the morning of Day 4, the Day of Discharge examinations will be conducted. After the time of discharge,

Philip Morris Products S.A. ZRHR-PK-02-JP

Clinical Study Protocol Final 1.0 / 21 June 2013 Confidential


subjects will then enter a 7-day safety follow-up (until Day 11) for the recording of spontaneously reported new AEs/SAEs and the active follow-up of ongoing AEs/SAEs.

### 4.4 Appropriateness of Measurement

All laboratory measures utilized for this study are validated and are appropriate for the study assessments.

All used questionnaires, except the cough questionnaire, are either available as a validated questionnaire in the local language or will be forward-translated and back-translated with subsequent independent verification.


#### 5 STUDY POPULATION

### 5.1 Selection of Study Population

Sixty-two Japanese female or male smoking healthy adult subjects, who smoke at least 10 CC per day, will be randomized into this study. The maximum number of CC is not limited. Subjects must have a smoking history of at least 3 years of consecutive smoking prior to Screening. The smoking status of the subjects will be verified based on a urine cotinine test (cotinine  $\geq$ 200 ng/mL).

#### 5.1.1 Inclusion Criteria

| | Inclusion Criteria | Rationale | Screening | Day of<br>Admission<br>(Day -1) |
|---|---|---|---|---|
| 1. | Subject has signed the ICF and is able to understand the information provided in the Subject Information Sheet and ICF. | Administrative | X | |
| 2. | Subject is aged from 23 to 65 years (inclusive). | Safety | X | |
| 3. | Subject is Japanese. | Effect | X | |
| 4. | Smoking, healthy subject as judged by the Investigator based on all available assessments in the Screening period/day of Admission (e.g., safety laboratory, spirometry [forced expiratory volume in 1 second {FEV <sub>1</sub> }/forced vital capacity {FVC} >0.7 at post-bronchodilator basal spirometry, post-bronchodilator FEV <sub>1</sub> >80% predicted value, and post-bronchodilator FVC >0.8], vital signs, physical examination, ECG, chest X-ray and medical history). | Safety | X | X |

Clinical Study Protocol Final 1.0 / 21 June 2013 Confidential


| | Inclusion Criteria | Rationale | Screening | Day of<br>Admission<br>(Day -1) |
|---|---|---|---|---|
| 5. | Subject smokes at least 10 commercially available CCs per day (no brand restrictions) with a maximum yield of 1 mg nicotine ISO/CC, as labeled on the cigarette package, for the last 4 weeks, based on self-reporting. Furthermore, the subject has been smoking for at least the last 3consecutive years. The smoking status will be verified based on a urinary cotinine test (cotinine ≥200 ng/mL). | Effect | X | X |
| 6. | The subject does not plan to quit smoking in the next 3 months. | Safety | X | |
| 7. | The subject is ready to accept interruptions of smoking for up to 4 days. | Safety | Х | X |
| 8. | The subject is ready to accept using both the THS 2.2 and NRT gum products. | Effect | | X |

### 5.1.2 Exclusion Criteria

Subjects who meet any of the following exclusion criteria must not be enrolled into the study:

| Exclusion Criteria | Rationale | Screening | Day of<br>Admission<br>(Day -1) |
|---|---|---|---|
| 1. As per Investigator judgment, the subject cannot participate in the study for any reason (e.g., medical, psychiatric, and/or social reason). | Safety | X | X |

Clinical Study Protocol Final 1.0 / 21 June 2013 Confidential


| | Exclusion Criteria | Rationale | Screening | Day of<br>Admission<br>(Day -1) |
|---|---|---|---|---|
| 2. | A subject who is legally incompetent, physically or mentally incapable of giving consent (e.g., emergency situation, under guardianship, prisoners or subjects who are involuntarily incarcerated). | Administrative | X | |
| 3. | The subject has medical condition requiring smoking cessation, or clinically relevant diseases (including but not limited to gastrointestinal, renal, hepatic, neurological, haematological, endocrine, oncological, urological, immunological, pulmonary and cardiovascular disease or any other medical condition [including but not limited to clinically relevant abnormal laboratory parameters]) in the judgment of the Investigator. | Safety | X | X |
| 4. | The subject has a body mass index (BMI) $<18.5$ or $\ge 32.0$ kg/m <sup>2</sup> . | Safety | X | X |
| 5. | As per Investigator judgment, the subject has medical conditions which require or will require in the course of the study, a medical intervention (e.g., start of treatment, surgery, hospitalization) which may interfere with the study participation and/or study results. | Effect | X | X |


| | Exclusion Criteria | Rationale | Screening | Day of<br>Admission<br>(Day -1) |
|---|---|---|---|---|
| 6. | The subject has used nicotine-containing products other than commercially available CC (either tobacco-based products or nicotine-replacement therapy) as well as electronic cigarettes and similar devices, within 4 weeks prior to assessment. | Effect | X | X |
| 7. | The subject has received medication (prescription or over-the-counter) within 14 days or within 5 half-lives of the drug prior to the Admission Day (Day -1; whichever is longer) that has an impact on CYP2A6 activity. | Effect | | X |
| 8. | In case the subject received any medication (prescribed or over-the-counter) within 14 days prior to Screening or prior to the Admission Day (Day -1) it will be decided at the discretion of the Investigator if these can potentially interfere with the study objectives and subject's safety. | Effect | X | X |
| 9. | The subject has a positive alcohol test and/or the subject has a history of alcohol abuse that could interfere with subject's participation in study. | Administrative | X | X |
| 10 | The subject has a positive urine drug test. | Administrative | X | X |
| 11 | Positive serology test for human immunodeficiency virus (HIV) 1/2, Hepatitis B or Hepatitis C. | Safety | X | |


| Exclusion Criteria | Rationale | Screening | Day of<br>Admission<br>(Day -1) |
|---|---|---|---|
| 12. Donation or receipt of whole blood or blood products within 3 months prior to Admission. | Safety | X | X |
| 13. The subject is a current or former employee of the tobacco industry or of their first-degree relatives (parent, sibling, child). | Administrative | X | |
| 14. The subject is an employee of the investigational site or any other parties involved in the study or of their first-degree relatives (parent, sibling, child). | Administrative | X | |
| 15. The subject has participated in a clinical study within 3 months prior to the Screening Visit. | Safety | X | |
| 16. The subject has previously participated in the same study at a different time (i.e., each subject can be included in the study population only once). | Administrative | X | |
| 17. For women only: Subject is pregnant (does not have negative pregnancy tests at Screening and at Admission) or is breast feeding. | Safety | X | X |
| 18. For women only: Subject does not agree to use an acceptable method of effective contraception.* | Safety | X | X |


\* Intrauterine device, intrauterine system, barrier methods of contraception (condoms, occlusive caps) with spermicidal foam/gel/film/suppository, hormonal contraception containing progesterone only, vasectomized partner(s) or true abstinence (periodic abstinence and withdrawal are not effective methods) from Screening until the end of the safety followup period. Hormonal contraception with estrogen containing products is NOT allowed in this study.

#### 5.1.3 Removal of Subjects from the Study

Subjects will be informed that they are free to withdraw from the study at any time. Subjects should be questioned for the reason of premature withdrawal, although they are not obliged to disclose it. This needs to be fully documented in the Source Document and electronic Case Report Form (eCRF).

When a subject withdraws or is removed from the study, the whole examination procedure planned on Day 4 must be performed as soon as possible after the time of withdrawal unless the subject has withdrawn their informed consent to do so. After the time of withdrawal, the subject will enter into the 7-day period of safety follow-up. Subjects withdrawn or removed from the study cannot re-enter the study.

Subjects must be withdrawn from the study for any of the following reasons:

- Withdrawal of informed consent.
- Any AE or condition (including clinically relevant changes in a laboratory parameter), at the discretion of the Investigator.
- Positive pregnancy testing (any invasive procedures, including the drawing of blood MUST NOT be performed after diagnosis of pregnancy, see Section 8.5.1.
- The Sponsor or Principal Investigator terminates the study. If the Sponsor or the Principal Investigator decide to prematurely terminates the study, the head of the medical institution should be reported the fact and the reason in writing promptly.
- Withdrawal is considered to be in the best interest of the subject or the other subjects.

Subjects may be discontinued from the study for any of the following reasons:

- Lost to follow-up.
- Concomitant treatment with non-authorized medication as defined in the context of this study (in general, any concomitant medication should be discussed with the Contract Research Organization (CRO) Medical Monitor on an ongoing basis).

Clinical Study Protocol Final 1.0 / 21 June 2013 

- If a subject uses any CC or nicotine/tobacco-containing product other than the product/regimen he/she is assigned to, it will be at the discretion of the Investigator to decide whether or not to withdraw the subject from the study.
- Non-compliance to the study procedures.

Subjects withdrawn prematurely after randomization will not be replaced and will not be allowed to re-enter the study. All subject withdrawals have to be documented properly in the source documentation and the eCRF.

#### 5.1.4 Violation of Selection Criteria

Subjects who are eligible at Screening, but who do not meet the entry criteria at Admission Day (Day -1) will be considered a screening failure and will be replaced by other subjects.

Subjects who violate the entry criteria prior to enrolment, but who were considered eligible, will be immediately withdrawn from the study when the violation is detected. If subjects are not yet randomized, they can be replaced.

ZRHR-PK-02-JP

Clinical Study Protocol Final 1.0 / 21 June 2013


#### INVESTIGATIONAL PRODUCTS AND REFERENCE POINT 6 **PRODUCT**

#### 6.1 Description

#### 611 **Investigational Products**

#### THS 2.2:

THS 2.2 comprises the following components: Tobacco Stick, Holder, Charger, a Cleaning Tool, a mains power supply, and a USB cable:

Charger: The function of the Charger (Model 4) is to recharge the Holder

after use. It contains a battery with sufficient capacity to recharge the Holder approximately 20 times. It is a convenient size to carry around, and can itself be recharged from a mains power source.

Tobacco Stick: The function of the Holder (Model 4.2) is to heat the Tobacco

Stick, delivering an aerosol to the user. The electrical heating is

Holder (Holder): powered from an internal battery which delivers power for about

6 minutes (allowing complete use of a single Tobacco Stick)

THS Tobacco Stick

The Tobacco Stick (product code C3) contains tobacco which, when heated, generates an aerosol. It is custom-designed to be used (Tobacco Sticks):

with the Holder.

The overall objective of the design is to provide an acceptable experience in which the HPHCs level in the aerosol is substantially reduced in comparison with CCs.

The THS 2.2 will be provided by the Sponsor.

Per cigarette/Tobacco Stick tar, nicotine, and carbon monoxide yields are normally determined by standardized test methods. The most widely used test method is ISO 4387. PMI has developed a modified version of this method, which improves the determination of tar in products with high water content, which is typical for heated tobacco products (PMI, 2012PMI, 2013a; PMI, 2013c). Another method is the more intensive smoking method developed by Health Canada (Health Canada, 1999).

| Philip Morris Products S.A. |
|-----------------------------|
| ZRHR-PK-02-JP |


Table 1 below lists the commonly reported measures:

Table 1 Measured aerosol fractions for the THS Tobacco Sticks

| Constituent (mg/THS Tobacco Stick) | ISO 1 | Health Canada Intense regime <sup>2</sup> |
|---|---|---|
| Tar/NFDPM | 4 | 10.3 |
| Nicotine | 0.5 | 1.32 |
| Carbon monoxide | 1 | 0.6 |

International Organization for Standardization ISO machine-smoking regimen. The analytical method has been modified to avoid inaccuracies as a result of condensation from high water-content aerosols.

#### **Reference Product:**

In the study sequences 1 and 2, the reference product to THS 2.2 is commercially available single brand CC with a maximum yield of 1 mg nicotine ISO per cigarette.

CC will not be provided by the Sponsor. All eligible subjects will be asked to purchase their own preferred single-brand CC prior to Admission. As randomization takes place on Day 0, every study subject needs to buy his/her anticipated amount of single-brand CC for a total of 2 days plus 2 extra packs.

#### 6.1.2 Reference Point Product

Nicotine replacement therapy gum (Nicorette® 2 mg gum) is the reference point product to THS 2.2 for sequences 3 and 4. The NRT gum will be supplied by the site and reimbursed by the Sponsor.

## 6.1.3 Packaging and Labeling

At Admission on Day -1, all study subjects will provide the anticipated amount of CC in sealed packs to the site staff. The cigarette packs provided by the subject should not be opened and the cellophane wrapper should be intact.

Each pack of cigarettes provided by the subject will be labeled to identify which subject the cigarettes belong to (labels should be affixed by the study site trial collaborator to the cellophane wrapper of the lower part of the pack). Packs of CC will be labeled to identify necessary information to match the subject with his/her suppliers.

Health Canada Intense machine-smoking regimen (55 mL puff volume, 2-second puff duration, 30-second inter-puff interval) (Health Canada, 1999)

Philip Morris Products S.A.

ZRHR-PK-02-JP

Clinical Study Protocol Final 1.0 / 21 June 2013 

For the Tobacco Sticks, the packs and cartons will be pre-labeled with the necessary information including but not limited to product code. The labels will be written in Japanese (Appendix 4).


### 6.2 Use of Investigational and Reference Point Products

Subjects will never be requested or forced to smoke and will be free to stop smoking at any time during the study. Subjects caught using any nicotine/tobacco product which is different from the assigned product will be withdrawn from the study. During the Screening period, subjects will be allowed to smoke according to their smoking habits except during the procedures of the Screening Visit (see Section 6.2) at the discretion of the site.

#### 6.2.1 Admission (Day -1)

Subject will be instructed not to smoke in the morning prior to Admission. Smoking *ad libitum* will be allowed throughout the day of admission except during the procedures until 11:00 PM. All subjects will be allowed to continue smoking *ad libitum* their preferred CC. All subjects (except women with a positive pregnancy test at Screening or Admission) will undergo a THS 2.2 test first (using up to 3 Tobacco Sticks) and subsequently NRT gum test at Day -1 prior to enrolment. Each subject will chew slowly the 2 mg NRT gum for 35±5 minutes while spacing each chew, leading to an administered dose of 1 mg nicotine/product use as per label similarly to the day of single use.

Following agreement that the THS 2.2 and NRT gum is acceptable, subjects will be enrolled and further randomized to 1 of 4 treatment sequences using an Interactive Web/Voice Response System.

#### 6.2.2 Investigational Period (Day 0 to Day 3)

During the first washout, each subject will maintain nicotine abstinence from Day -1 at 11:00 PM to the time of single use of his/her allocated product at Day 1. At Day 1, after the single use of the product, subjects will maintain nicotine abstinence for the rest of the day. During the second washout on Day 2, subjects will maintain nicotine abstinence until the time of single use of subject's allocated product at Day 3. Subjects will not be allowed to smoke or use any other nicotine/tobacco-containing products other than the products/regimen they are allocated to.

Time point of first product use during study day  $(T_0)$  will be defined as start of the single product use at the single use days. The start time of the use of each product has to be documented on single use days (Day 1 and Day 3). The start of product use for THS 2.2 is defined as the time of the first puff. The start time for CC corresponds to the lighting of the CC, and the start time of the NRT gum is the time of the NRT gum intake. The 30 seconds it takes to pre-heat the Holder will not be taken into account. The subject must not take a puff of the Tobacco Stick during the pre-heating time.


For NRT gum, the start time and the stop time will be documented in appropriate log.

The start of the first product use can be different for each subject both days of product use; however, it must be in the window of 6:00 AM to 9:00 AM.

### Single use of products (Day 1 and Day 3):

On Day 1 and Day 3, subjects will use the product they are randomized to only once in the morning between 6:00 AM to 9:00 AM, and will abstain from the product or other nicotine/tobacco-containing items for the rest of the day, i.e., subjects in the THS 2.2 arm will use one Tobacco Stick, subjects in the CC arm will smoke one CC, and subjects in the NRT gum arm will chew slowly the 2 mg NRT gum for 35±5minutes while spacing each chew (leading to an administered dose of 1 mg nicotine/product use as per label

| | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 |
|-------|------------|------------|------------|------------|
| Day 1 | THS 2.2 | CC | THS 2.2 | NRT gum |
| Day 3 | CC | THS 2.2 | NRT gum | THS 2.2 |

#### 6.2.3 Day of Discharge/Time of Discharge

On the Day of Discharge (Day 4), smoking will be only allowed after all laboratory procedures and the spirometry have been performed. All examinations of the Day of Discharge will be conducted on Day 4 prior to the time of Discharge.

### 6.2.4 Safety Period

During the safety follow-up period, subjects are free to smoke according to their usual smoking habits.

#### 6.2.5 Stopping Rules for Investigational Product

For safety purposes, smoking the THS 2.2 or the CC or the use of the NRT gum should be temporarily stopped in the event of any signs suggesting nicotine overexposure, e.g., gastrointestinal disturbance (nausea, vomiting, diarrhea, stomach, or abdominal pain), cold sweats, headache, dizziness and breathing problems, or any reasons at the discretion of the Investigator.


### 6.3 Method for Assigning Subjects to Study Arms

Randomization to product exposure sequence will be done through an Interactive Telephone and Web Response System.

Each sex and each of the smoking level (ISO nicotine levels  $\le$ 0.6 mg and >0.6 to  $\le$ 1 mg) will have a quota applied to ensure they represent at least 40% of the total study population allocated within each of the following analysis groups:

- Group 1: composed of sequences 1 and 2.
- Group 2: composed of sequences 3 and 4.

In particular, the maximum number of subjects having the same sex or nicotine level value will be limited to 26 in Group 1 and 10 in Group 2.

The randomization of the planned sample size of 62 subjects will be ensured by applying quota to the number of subjects per each sequence (22 subjects for sequences in Group-1, and 9 subjects for sequences in Group-2).

Subjects will be randomly assigned to one of the four product exposure sequences by means of a permuted-block schema. Block size and other randomization details will be available in the randomization plan.

The randomization plan will be generated by an independent statistician and none of the Sponsor staff, Investigators or study subjects will have access to the randomization schema prior to randomization.

## 6.4 Blinding

This is an open-label study; therefore the subjects and investigators will be unblinded to subject's sequence. However, there will be a limited degree of blinding in the data review and data analysis process. In particular, PMI and CRO personnel will be blinded to the randomized sequence as summarized in the following table:

| Blinded Study Personnel | End of Blinding Period |
|---|---|
| PMI and CRO study statisticians | After the Statistical Analysis Plan (SAP) finalization or PMI blind database review <sup>(*)</sup> , whichever comes last. |
| PMI data manager | After the finalization of PMI blind database review. (*) |

| Philip Morris Products S.A. | Clinical Study Protocol | Confidential |
|---|---|---|
| ZRHR-PK-02-JP | Final 1.0 / 21 June 2013 | |
| PMI safety and clinical scientist | After the finalization of PMI blind<br>be actively un-blinded before that to<br>occurrence of any safety question, v | time point in case of the |

(\*) As part of the PMI Quality Control (QC) activity, data listings will be reviewed by PMI before database lock, with no access to the randomization sequence information

Any PMI and CRO personnel who are not listed in the above table will be unblinded by default.

## 6.5 Investigational Product Accountability and Compliance

### 6.5.1 Dispensing Investigational Product and Reference Point Products

From Day -1 until Day 4, the THS 2.2, NRT gum, and CC will be dispensed by the Investigators or dedicated study collaborator, as per study design. Each dispense of the product will be recorded in a log. The log should include subject number, date and start time of product use. The product will not be promoted for commercial distribution or test market.

#### 6.5.2 Storage and Accountability

The THS 2.2, NRT gum and CC will be stored in a secured site storage place with access limited to the authorized personnel only. Full accountability of the distributed products will be ensured by designated collaborator. Subjects will return each butt of any used Tobacco Stick or CC immediately after use to the site study collaborator for accountability. They will also return each used NRT gum after use to the site study collaborator. This will be documented in appropriate log. On the time of discharge, unused CCs given to the site staff at Admission on Day -1 will be given back to the subjects.

#### 6.5.3 Investigational Product Retention

Unused Tobacco Sticks and NRT gum will be destroyed if possible, or returned to the Sponsor upon study completion. The Tobacco Heating Devices will be returned to the Sponsor.

### 6.5.4 Compliance to Investigational Products

Compliance for all arms will be ensured by strict distribution of the products (product by product) and collection of used Tobacco Sticks, the CC butts and the NRT gum after use will be documented in appropriate logs.


In addition, for subjects using NRT gum, the compliance will be chemically verified using exhaled CO breath. The cut-off point for the CO breath test value to distinguish tobacco use vs. no tobacco use will be 10 ppm (Benowitz et al., 2002).

Furthermore, the CO breath test will be considered as one of the measures of compliance during the wash-out days in all subjects.

#### 6.6 Restrictions

### 6.6.1 Smoking Restrictions

On Day 1 and Day 3, to avoid nicotine cross contamination, users of THS 2.2 and smokers of CC will use or smoke, as applicable, in dedicated separate rooms: one room for THS 2.2 and one room for CC. Every subject must use or smoke, as applicable alone with an interval between subjects allowing ventilation of the room. Subjects receiving NRT gum must not have access to these rooms.

In the morning prior admission, subjects will be instructed not to smoke. At admission, smoking is only allowed during the designated smoking times from 6:30 AM to 11:00 PM as detailed in the study design. Subjects will not have free access to their NRT gum, CC or THS 2.2, which will be dispensed by the site staff individually as described in Section 6.5.1.

Smoking is not allowed during study procedures except during blood sampling for nicotine PK on Day 1 and Day 3. Furthermore, smoking is not allowed on Day 4 until all laboratory tests and the spirometry have been conducted.

During the days of wash-out or single product use (for CC and THS 2.2 arms), no NRT gum or other products supportive to SA must be used or will be provided to the subjects.

#### 6.6.2 Dietary Restrictions

A standard diet will be designed by a dietician for the whole confinement period. For each meal, the caloric and fat content should be controlled in order to avoid a "high-fat" diet. The FDA guidance on food-effect studies for bioequivalency testing identifies a "high-fat" diet as a diet which maintains approximately 50 percent of total caloric content of the meal and is high in calories (approximately 800 to 1000 calories) (FDA, 2002).

Subjects are not allowed to bring their own food or beverages to the investigational site. Meals will be served according to the schedules provided in Section 9. Additional light snack, fruits, and raw vegetables can be distributed to the subjects without restrictions at any time during confinement as long as they fulfill the above requirements described in this section. Consumption of water is allowed as desired. The same menu and meal schedule will be administered uniformly for all subjects in all study arms. Fasting state has to be observed

Clinical Study Protocol Final 1.0 / 21 June 2013 

for at least 10 hours prior to blood draws for the safety laboratory at the Screening Visit, on Day -1, and Day 4.

#### 6.6.3 Concomitant Medication

For the purpose of this study, no concomitant medication should be taken by the subjects. Any medication with an impact on the CYP2A6 metabolism (as prescription and over-the-counter products) as given below must be avoided as CYP2A6 is involved in the nicotine metabolism (see Table 2).

In this study the use of hormonal contraception containing estrogens is NOT allowed. This also applies to hormone replacement therapy. Only hormonal contraception with products containing progesterone is allowed during this study. Subjects using estrogens during the study will be withdrawn.

The following drugs and substances are considered as having an impact on CYP2A6 activity (Lacy et al., 2007). Prior to database close, the concomitant medication will be assessed according to the potential impact on CYP2A6 activity and the potential impact on study results.


### Table 2 Drugs and Substances Considered Interacting with CYP2A6

| Drug name | Substance Class |
|---|---|
| Fluoroquinolones, including ciprofloxacin and ofloxacin, nafcillin, rifampicin | Antibiotic |
| Fluvoxamine, fluoxetine, paroxetine, bupropion, duloxetine, amitriptyline, imipramine, sertraline, mirtazapine, citalopram, thioridazine | Antidepressant |
| Haloperidol, perphenazine, chlorpromazine, propoxyphene fluphenazine, clozapine, olanzapine | Neuroleptic |
| Phenobarbital, primidone, carbamazepine | Antiepileptic |
| Cholorquine, quinidine | Antirheumatic |
| Clotrimazole, terbinafine, fluconazole, ketoconazole, miconazole | Antimycotic |
| Erythromycin, ciprofloxacin, clarithromycin, norfloxacin | Antibiotic |
| Cimetidine, chlorpheniramine, diphenhydramine, ranitidine | H2-receptor antagonist |
| Amiodarone, verapamil, mibefradil, mexiletin, propafenone, propranolol, lidocaine | Antiarrhythmic |
| Losartan, amlodipine, nifedipine | Antihypertensive |
| Drospirenone, estrogens | Hormonal contraceptives |
| | Agents for hormonal replacement therapy (estrogens) |
| Fluvastatin | Cholesterol-lowering agent |
| Theophylline | Antispasmodic pulmonological agent/Bronchodilator agent |
| Omeprazole, Lansoprazole | Proton pump inhibitor |
| Interferon | Antiviral/Immunomodulating agent |
| Methoxsalen | Anti-psoriatic (substance class<br>Furocoumarins) |

Clinical Study Protocol Final 1.0 / 21 June 2013


| Modafinil, Diclofenac, Rofecoxib | Analgesic |
|---|---|
| Insulin | Anti-diabetic |
| Sildenafil | Phosphodiesterase-Inhibitor (e.g., used for treatment of Erectile dysfunction) |
| Quinine | Crystalline alkaloid |
| St. John's Wort | Over-the-counter (herbal remedy) antidepressant |
| Psoralen | Anti-psoriatic (substance class<br>Furocoumarins) |
| Pilocapine | Cholinergic agonists (e.g., used for Glaucoma Therapy) |

Data source: Lacy et al., 2007. This list is not exhaustive.

However, the Principal Investigator is responsible for the medical care of the subjects during their participation in this study. Any decisions regarding the prescription of medication will be taken in the best interest of the subject.

If the use of a concomitant medication cannot be avoided for the subject's safety it has to be fully documented (for details, see Section 7.4.5) Concomitant medications should be followed up with the CRO Medical Monitor on an ongoing basis.

Concomitant medication will first be assessed at Screening Visit. To be eligible for the study any medication with impact on CYP2A6 metabolism must be discontinued at least 14 days prior to Admission to the clinic or for at least five half-lives (whichever is longer). They must not be used during the entire study until the time of discharge. It is at the discretion of the Investigator to assess if a termination of such medication at Screening is medically justified and safe for the subject.

#### 6.6.4 Others

From admission to discharge, practice of intensive exercise and physical work-out will be prohibited as it may impact nicotine absorption profile.


#### 7 STUDY PROCEDURES

Personnel performing study measurements or recording must have the appropriate training fully documented. Quality control (QC) measures have to be in place. All study procedures are provided as an overview in the Schedule of Events (Appendix 1). In this Section, only the expected/planned time points for the various measurements are given. Considering that not all subjects can have a procedure at the same time point, adequate time windows will be given for each study procedure and each time point in Section 9. Site study collaborator will adhere to the site's Standard Operating Procedures (SOPs) for all activities. Appropriate medical advice will be provided to the subject in case of any medical findings requiring health care.

#### 7.1 Informed Consent

Each subject must give his/her informed consent prior to participating in the study. During the consent process, the Investigator obtaining consent must inform each subject of the nature, risks, benefits of and alternatives to study participation. In addition, each subject must have sufficient time to review the ICF in order to understand it, and have adequate opportunity to ask questions. The ICF must be signed and dated by the subject prior to any study-specific procedures taking place.

## 7.2 Smoking Cessation Advice and Debriefing

Each subject will be given advice on the risks of smoking 3 times during the study: at the Screening Visit, at Admission (Day -1), and at Day 4. This will take the form of a brief interview according to WHO recommendations (WHO, 2002). Details of the interview will be recorded in the Source Document File. Information on the risk of smoking will be given to the subjects on an individual basis during a face-to-face meeting between the subject and the Investigator, and may additionally be given in a group session.

In addition to the smoking cessation advice, a debriefing of subjects will be done at each smoking cessation advice session to address any intended or unintended beliefs participants have about the candidate MRTP. The goal of the debriefing would be to help ensure that subjects exit the study with an accurate understanding of product risks, including an understanding that the candidate MRTP has not been demonstrated to be less harmful.


## 7.3 Support during Smoking Abstinence/Periods of Reduced Smoking

All subjects will be closely monitored by the site staff on Day 0, Day 1; Day 2, and Day 3. This includes monitoring of clinical tests e.g., vital signs, physical examination, and body weight. It also refers to close monitoring of the subject's behavior, AEs, and his/her mood.

#### 7.4 Clinical Assessments

Any clinically relevant finding detected during the Screening Visit has to be documented as a concomitant disease. This also applies to clinically relevant findings (e.g., laboratory values, vital signs and ECGs) detected during the Screening Visit. Any untoward medical occurrence in a subject detected during the study which was not present at the Screening Visit must be documented as an AE. Worsening of a pre-existing condition from the Screening Visit onwards will also be documented as an AE. If a clinically relevant finding is detected during the Screening period, the Investigator needs to check if inclusion criterion no. 4 is still fulfilled

### 7.4.1 Demographic Data

Demographic data (sex, date of birth/age) will be recorded at the Screening Visit.

### 7.4.2 Identification of the Current Cigarette Brand

Identification of the current CC brand(s) smoked by the subject will be done at the Screening Visit and at Day -1. At the Screening Visit, smokers will be asked to bring a pack of their current CC brand(s) to the site. On Day -1, subjects will hand their CC supply for the entire confinement period to the site study collaborator. The site study collaborator will document the brand name and yields. A photograph of the front and the side of the cigarette pack supplied by the subject (bearing the tar, and nicotine yields) will be taken by the study site staff in addition to recording the brand name and yields. These photographs will be considered as Source Documentation. A copy of the photographs will be provided to the Sponsor electronically (as Digital Video Disk or Compact Disc [CD]).

### 7.4.3 Smoking History and Willingness to Quit Smoking

Subjects will be questioned for their smoking history. At Screening and on the Day of Admission (Day -1) this will include questions to evaluate whether the subject has smoked for at least the last 3 consecutive years, to determine the number of CC smoked during the previous 4 weeks, and to evaluate if the CCs smoked during the previous 4 weeks were CCs. At the Screening Visit only, the subject will also be asked if he/she plans to quit smoking within the next 3 months. In addition, the subject will be asked if he/she has used nicotine-containing products other than commercially available CC (either tobacco-based products or


nicotine replacement therapy), electronic cigarettes or similar devices, within 4 weeks prior to assessment.

At Screening and on the Day of Admission (Day -1), subjects will also be asked if they are willing to abstain from smoking for at least 4 days (as required in the study protocol inclusion criteria). Only subjects who are prepared and able to comply with this requirement will be considered for participation in the study.

#### 7.4.4 Demonstration and Trial of the THS 2.2 and NRT Gum

All subjects will have a demonstration of the THS 2.2 product and the NRT gum at the Screening Visit by the study site collaborator. On Day -1 as last procedure of the eligibility assessments on that day, subjects will have a product test prior to enrolment, first THS 2.2 (use of up to 3 Tobacco Sticks) and subsequently NRT gum. Each subject will chew slowly the 2 mg NRT gum for 35±5 minutes while spacing each chew, leading to an administered dose of 1 mg nicotine/product use as per label similarly to the day of single use.

In female subjects, the THS 2.2 and NRT gum product tests must only be done after pregnancy is excluded by a urine pregnancy test. Only subjects willing and ready to use the THS 2.2 and NRT gum can be enrolled into the study.

### 7.4.5 Medical History, Concomitant Disease, Previous and Ongoing Medications

Relevant medical history and any concomitant disease will be documented at the Screening Visit. Medical history is defined as any condition that started prior to and ended prior to Screening. A concomitant disease is defined as any condition that started prior to the Screening Visit and is still ongoing at the Screening Visit.

Prior medication taken within 4 weeks prior to Screening Visit and any concomitant medication needs to be documented. Any medication which was started prior to the Screening Visit and is still being taken by the subject will be considered a concomitant medication. Medication initiated after Screening is also referred to as concomitant medication. This applies to both prescription and over-the-counter products.

Records of any medication taken must include the drug name (preferably both generic and trade name), route of administration (e.g., oral, intravenous), total daily dose/unit (e.g., expressed in mg, ml, or IU), indication, the start and (if applicable) the stop date (day, month, and year). Any therapy changes (including changes of regimen) during the study are to be documented. Any concomitant medication that is still being taken by the subject at EOS will be recorded on the eCRF.

Clinical Study Protocol Final 1.0 / 21 June 2013


#### 7.4.6 Physical Examination

A physical examination will be conducted at the Screening Visit, at Admission (Day -1), and at the Day of Discharge (Day 4).

#### 7.4.7 **Body Height and Weight**

Body weight will be recorded at the Screening Visit, at Admission (Day -1) and at the Day of Discharge (Day 4). Body height will be measured at the Screening Visit only. The BMI will be calculated from the body weight and height using the following formula, rounded to one decimal place:

$$BMI = \frac{\text{weight in kilograms}}{\text{height in meters}^2} = \frac{kg}{m^2}$$

#### 7.4.8 Vital Signs

Systolic and diastolic blood pressure, pulse rate, and respiratory rate will be measured at the Screening Visit, at Admission, and at every day in confinement. All parameters will be recorded in supine position after the subject has rested for at least 5 minutes.

For every measurement, it will be documented if the subject has smoked within 15 minutes prior to the measurement.

#### 7.4.9 Other Clinical Assessments

#### 7.4.9.1 Spirometry

Spirometry with and without a short-acting bronchodilator will be done at the Screening Visit to evaluate inclusion/exclusion criteria (the post-bronchodilator results). At screening, spirometry without bronchodilator will be done first, and then, spirometry with bronchodilator. Furthermore, spirometry without bronchodilator will be performed at Day -1 (baseline values) and at Day 4 (for comparison with the baseline values). Spirometry has to be done prior to smoking the first cigarette of the day.

Spirometry will follow the 2005 testing and quality recommendations by the American Thoracic Society/European Respiratory Society Joint Task Force on the standardization of spirometry along with the electronic data submission and documentation processes. Spirometry predicted values will be standardized to the NHANES III predicted set.

All personnel performing lung function testing should have the appropriate training and quality control (QC) measures should be put into place and be properly documented and filed

Clinical Study Protocol Final 1.0 / 21 June 2013 Confidential


at the pulmonary function laboratory (including the records of the calibration, if applicable). The  $FEV_1$  and FVC will be recorded.

The subject will be submitted to a spirometry with maximum voluntary ventilation measurement.

For spirometry, assessed parameters will include:

- FEV<sub>1.</sub>
- FVC.
- FEV<sub>1</sub>/FVC.

### 7.4.9.2 Electrocardiogram

An ECG will be recorded at Screening and on the following study days: Day 1 and Day 3. The ECG testing will be performed as per the site local practice. A standard 12-lead ECG will be recorded after the subject has rested for at least 10 minutes in supine position.

The following parameters will be documented: heart rate, PR interval, QRS interval, QT interval, and QTc interval corrected by the ECG device according to Bazett's formula. Every ECG has to be assessed as normal, abnormal – clinically not relevant, or abnormal – clinically relevant. A diagnosis has to be provided in the Case Report Form for all ECGs assessed as abnormal – clinically relevant. Electrocardiogram print-outs will be interpreted by a qualified physician. Any print-outs of ECGs on thermo-sensitive paper must be photocopied, initialed, dated and stapled together for inclusion in the Source Data File.

#### 7.4.9.3 Chest X-ray

A chest X-ray (anterior-posterior and left lateral views) will be assessed during the Screening period to exclude subjects with relevant pulmonary diseases. Subjects will be referred to a radiology facility for this procedure. No new examination is required if the subject can present a chest X-ray with anterior-posterior and left lateral views at the Screening Visit which is not older than 6 months.

#### 7.5 Biomarker Assessment

All bioanalytical assays and laboratory assessments (Section 7.6) will be carried out using validated methods. The bioanalytical methods used will be documented in the Bioanalytical Plans/Report. A list of laboratories is provided in Appendix 2.

Philip Morris Products S.A.

ZRHR-PK-02-JP

Clinical Study Protocol Final 1.0 / 21 June 2013 Confidential


The start time of the use of each product has to be documented on single use days (Day 1 and Day 3). For NRT gum specifically, the time of NRT gum use (start time  $T_0$ ), and the stop time of NRT gum use needs to be recorded.

Precautions should be taken during blood sampling and processing to prevent the contamination of samples with environmental nicotine or CO.

### 7.5.1 Biomarkers of Exposure

#### 7.5.1.1 Biomarkers of Exposure to CO and COHb

Carboxyhemoglobin measured in blood and exhaled CO will be investigated as a measure of exposure to CO. The CO breath test will also serve as a measure of compliance in subjects using NRT gum as well as on the wash-out days in all subjects.

#### CO Breath Test

CO in exhaled breath will be measured using the Smokerlyzer $^{\circledR}$  device such as Micro+TM Smokerlyzer $^{\circledR}$  deviceor similar . The test will be performed for all subjects including the subjects using the NRT gum.

A CO breath test will be conducted once on Day -1 and Day 4:

On Day 0, Day 1, Day 2, and Day 3, four CO breath tests will be done per day. On Day 1 and Day 3, the first test per day will be performed within 15 minutes prior to  $T_0$ . The three other tests will be conducted as described in section 9. On the wash-out days (Day 0 and Day 2), the first test will be conducted between 8:00 AM-9:30 AM the three other tests will be conducted as described in section 9

#### Carboxyhemoglobin

Tests for COHb measurement will be performed at a local laboratory.

Blood samples will be taken as follows at Day 1 and Day 3:

A total of 5 blood samples will be taken. The first sample will be taken within 15 minutes prior to using the first product  $(T_0)$ . Thereafter, the sampling times in relation to  $T_0$  are at 15 minutes, 60 minutes, 4 hours and 12 hours post- $T_0$ .

#### 7.5.1.2 Biomarkers of Exposure to Nicotine

Blood samples to measure nicotine in plasma will be taken as follows:

Clinical Study Protocol Final 1.0 / 21 June 2013


#### Single Use on Day 1 and Day 3 for THS 2.2 and CC only:

A total of 16 blood samples will be taken for a 24-hour profile (Day 1 and Day 3). The first blood sample will be taken within 15 minutes prior to the single use ( $T_0$ ). Times of sampling are thereafter in relation to  $T_0$ :  $T_1$  after 2 minutes,  $T_2$  after 4 minutes,  $T_3$  after 6 minutes,  $T_4$  after 8 minutes,  $T_5$  after 10 minutes,  $T_6$  after 15 minutes,  $T_7$  after 30 minutes,  $T_8$  after 45 minutes,  $T_9$  after 60 minutes,  $T_{10}$  after 2 hours,  $T_{11}$  after 4 hours,  $T_{12}$  after 6 hours,  $T_{13}$  after 9 hours,  $T_{14}$  after 12 hours and  $T_{15}$  after 24 hours (this sample will be drawn during the day following product use, i.e., wash-out).

### Single Use on Day 1 and Day 3 for NRT gum only:

A total of 16 blood samples will be taken for a 24-hour profile (Day 1 and Day 3). The first blood sample will be taken within 15 minutes prior to the single use ( $T_0$ : Times of sampling are thereafter in relation to  $T_0$ :  $T_1$  after 10 minutes,  $T_2$  after 20 minutes,  $T_3$  after 25 minutes,  $T_4$  after 30 minutes,  $T_5$  after 35 minutes;  $T_6$  after 40 minutes;  $T_7$  after 45 minutes,  $T_8$  after 60 minutes,  $T_9$  after 2 hours,  $T_{10}$  after 3 hours,  $T_{11}$  after 4 hours,  $T_{12}$  after 6 hours,  $T_{13}$  after 9 hours  $T_{14}$  after 12 hours and  $T_{15}$  after 24 hours (this sample will be drawn during the day following product use, i.e., wash-out).

#### 7.5.2 CYP2A6 Activity

CYP2A6 activity will be measured in plasma on Day -1. CYP2A6 activity drives the metabolism of nicotine to cotinine and subsequent metabolites. In this study the CYP2A6 activity will be measured using the metabolic molar ratio of *trans*-3'-hydroxycotinine/cotinine (Jacob et al., 2011).

## 7.6 Laboratory Assessments

A list of laboratories is provided in Appendix 2.

### 7.6.1 Clinical Chemistry, Hematology, and Urine Analysis for Safety Panel

Haematology, clinical chemistry and urine analysis for the safety panel will be measured at Screening, at Day of Admission (Day -1), and at the Day of Discharge (Day 4). Tests will be conducted at a local laboratory or the site. Blood will be taken after no less than the 10 hours of fasting (see Section 6.6.2). The urine test will be performed semi-quantitatively as urine test at the site. Parameters to be measured are listed in Table 3.


Table 3. Clinical Laboratory Parameters for Safety Panel

| Hematology | Clinical chemistry | Urine analysis |
|---|---|---|
| - Hematocrit | - Albumin | - pH |
| - Hemoglobin | - Total protein | - Bilirubin |
| - Mean corpuscular hemoglobin | - Alkaline phosphatase | - Glucose |
| - Mean corpuscular hemoglobin | - Alanine aminotransferase | - Nitrite |
| concentration | - Aspartate aminotransferase | - Red blood cell traces |
| - Mean corpuscular volume | - Blood urea nitrogen | - Protein |
| - Platelet count | - Creatinine | - Specific gravity |
| - Red blood cell count | - Gamma-glutamyl transferase | |
| - White blood cell (count) (WBC) | - Fasting glucose | |
| - Differential WBC count: | - Lactate dehydrogenase | |
| <ul> <li>Neutrophils</li> </ul> | - Potassium | |
| Basophils | - Sodium | |
| <ul> <li>Eosinophils</li> </ul> | - Total bilirubin | |
| <ul> <li>Lymphocytes</li> </ul> | - Direct bilirubin | |
| <ul> <li>Monocytes</li> </ul> | - Total cholesterol | |
| | - Triglycerides | |

### 7.6.2 Serology

A test for Hepatitis B surface antigen, Hepatitis C virus and HIV (anti-HIV1/2 and p24 antigen) will be done at Screening. In case of positive results, the subject will be referred to appropriate medical care.

### 7.6.3 Urine Drug Screen

A urine drug screen will be performed at the site at the Screening Visit and at the day of Admission. The urine will be screened for amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, and opiates.

#### 7.6.4 Urine Cotinine Screening

A urine cotinine test will be performed at Screening and at Admission to the clinic in order to confirm the subject's smoking status. The test must detect cotinine with a cotinine of  $\geq$ 200 ng/mL.

Clinical Study Protocol Final 1.0 / 21 June 2013


#### 7.6.5 Alcohol Breath Test

Subjects will undertake a breath alcohol test at the Screening Visit and at Admission to the clinic using a newly calibrated alcometer device.

#### 7.6.6 Urine Pregnancy Testing

All female subjects will undergo pregnancy testing at the Screening Visit, at Admission to the clinic, and at the Day of Discharge (Day 4). Female subjects with a positive pregnancy test at the Screening Visit or on Day -1 cannot be enrolled and are considered a screening failure. Pregnancy in such subjects will not be followed up as no exposure to the THS 2.2 will have occurred. Product test at Admission must be done only in female subjects with a negative pregnancy test. In any case of a positive pregnancy test, the Investigator will inform the subject about the risks associated with smoking during pregnancy. In the event of unclear urine pregnancy test in peri-menopausal women, absence of pregnancy should be confirmed by a serum follicle stimulating hormone level >20 IU/l.

All pregnancies detected during the study must be reported and handled as described in Section 8.5.1.

### 7.7 Sample Handling, Storage, and Shipment

All blood samples are to be tested at a central laboratory with the exception of COHb blood samples and the safety laboratory samples which will be tested at a local laboratory (see Appendix 2). The urine drug screen, urine pregnancy tests and urine cotinine tests will be done by the site study collaborator at the site. The tests will be provided by the sites.

Detailed procedures for handling of samples are described in the separate sample handling manual (SHM). Safety laboratory samples will be destroyed as by the laboratories standard procedures. All other samples will be destroyed once the Clinical Study Report (CSR) has been finalized. The facility/-ies at which the samples are stored will be informed in writing by the Sponsor when destruction of the samples shall be performed.

#### 7.7.1 Blood samples

Blood samples will be drawn by qualified and trained site personnel. Subjects should be in a seated position during blood collection. The maximal total volume of blood drawn for each subject will be around 190 mL. The required aliquots and volumes for assessments of blood/plasma parameters and tests are summarized in the SHM.

Clinical Study Protocol Final 1.0 / 21 June 2013


### 7.7.2 Urine samples

Spot urine samples will be taken for urine drug screen, cotinine screen, pregnancy tests and safety urinalysis.

#### 7.8 Questionnaires

The subject questionnaires and the Visual Analogue Scale (VAS) will be entered by the subject directly in the electronic patient reported outcomes (ePRO) device. The questionnaires and the VAS will be reviewed for completeness by the study site collaborator and subjects will be requested to complete any missing information.

Symptoms or worsening of symptoms as documented on any of the questionnaires or the VAS do not need to be documented as AEs because the questionnaire and the VAS will be analyzed as part of the report. However, it is at the discretion of the Investigator to document such symptoms also as AEs. The main source for AE collection will be the face-to-face interview between the subject and the study site collaborator using, open, non-directive questions (see Section 8.2.1).

### 7.8.1 Fagerström Test for Nicotine Dependence (revised version)

Potential nicotine dependence will be assessed at Screening using the FTND in its revised version (Fagerström and Schneider, 1989), as updated in 2012 (Fagerström et al., 2012).

The questionnaire consists of 6 questions which have to be answered by the subject himself/herself. The scores obtained on the test permit the classification of nicotine dependence into three levels: Mild (0 to 3 points); Moderate (4 to 6 points); Severe (7 to 10 points) (Fagerström et al., 2012).

#### 7.8.2 Assessment of Cough

Subjects will be asked if they have experienced a regular need to cough e.g., coughing several times in the last 24 hours prior to assessment. If the answer is 'yes', they will be asked to complete a VAS, 3 Likert scales and an open question also assessing the previous 24 hours. The questionnaire will be asked prior to product use.

The VAS will assess how bothersome cough is to the subject ranging from 'not bothering me at all' to 'extremely bothersome'.

Furthermore, subjects will be asked to assess the intensity and frequency of cough and the amount of sputum production on Likert scales:


- The intensity of cough will be assessed on a 5-point Likert scale ranging from 1 to 5: 1 = very mild; 2 = mild; 3 = moderate; 4 = severe; 5 = very severe.
- The frequency of cough will be assessed on a 5-point Likert scale ranging from 1 to 5: 1 = rarely; 2 = sometimes; 3 = fairly often; 4 = often; 5 = almost always.
- The amount of sputum production will be assessed on a 4-point Likert scale ranging from 0 to 3: 0 = no sputum; 1 = a moderate amount of sputum; 2 = a larger amount of sputum; 3 = a very large amount of sputum.

Finally, subjects will be asked with an open question if there are any other important observations that they would like to share with the staff about their coughing.

Assessments will be done on a daily basis from Day 0 to Day 4. On Day 2 and Day 4, questionnaire must be asked 24 hours after T<sub>0</sub> of Day 1 and after 24 hours after T<sub>0</sub> of Day 3.

### 7.8.3 Modified Cigarette Evaluation Questionnaire (modified version)

Product evaluation will be assessed using the MCEQ (Cappelleri et al., 2007). The MCEQ assesses the degree to which subjects experience the reinforcing effects of smoking, by measuring:

- Smoking satisfaction (satisfying, tastes good, enjoy smoking).
- Psychological rewards (calms down, more awake, less irritable, helps concentrate, reduces hunger).
- Aversion (dizziness, nauseous).
- Enjoyment of respiratory tract sensations (single-item assessment).
- Craving reduction (single-item assessment).

This questionnaire will only be completed by the subjects who use the THS 2.2 or smoke CC during the study in sequence 1 and 2. The MCEQ will be completed by subjects on Day 1 and Day 3.

### 7.8.4 Questionnaire of Smoking Urges brief

To assess the urge-to-smoke, all subjects will be asked to complete a 10-item brief version of the QSU-brief (Tiffany et al., 1991). The QSU-brief is a self-reported questionnaire with 10 items to be rated on a 7-point scale, ranging from 1 (strongly disagree) to 7 (strongly agree). Higher scores in this questionnaire indicate a higher urge to smoke.

The findings in this brief version were consistent with the expressions of craving found in the 32-item version of the QSU-brief (Tiffany et al., 1991). The findings supported a Confidentiality statement: Data and information contained in this document are considered to constitute trade secrets and confidential commercial information, and the legal protections provided to such trade secrets and confidential information are hereby claimed under the provisions of applicable law. No part of this document may be publicly disclosed without the written consent of Philip Morris Products S.A.

Philip Morris Products S.A.

ZRHR-PK-02-JP

Clinical Study Protocol Final 1.0 / 21 June 2013 Confidential


multi-dimensional conceptualization of craving to smoke and demonstrated the utility of a brief multi-dimensional measure of craving (Cox et al., 2001).

The QSU-brief will be completed by the subject himself/herself at single use study days.

#### 7.8.4.1 THS 2.2 and CC arms QSU-timing:

For subject on THS 2.2 or on CC: first sample within 15 min prior to  $T_0$ , 9 assessments thereafter in relation to  $T_0$ : 15 min, 30 min, 45 min, 60 min, 2 hr, 4 hrs, 6 hrs, 9 hrs, and 12 hrs after  $T_0$ .

#### 7.8.4.2 NRT gum arm QSU-timing:

For subjects on NRT gum: first sample within 15 min prior to  $T_0$ , 9 assessments thereafter in relation to  $T_0$ : 20 min, 30 min, 45 min, 60 min, 2 hr, 4 hr, 6 hrs, 9 hrs, and 12 hrs after  $T_0$ .


### 8 ADVERSE EVENTS

#### 8.1 Definitions

#### 8.1.1 Adverse Events

The FDA MRTP guidelines specify the following definition for AEs for tobacco products FDA, 2012a:An AE is any health-related event associated with the use of a tobacco product in humans, which is adverse or unfavorable, whether or not it is considered related to the tobacco product, as defined by the MRTP guidelines.

An AE is defined as any untoward medical occurrence in a subject, or clinical investigation subject administered an IP, which does not necessarily have a causal relationship with the IP or reference point product. An AE can therefore be any unfavorable and unintended sign (including a clinically relevant abnormal laboratory finding), symptom, or disease temporally associated with the use of an IP or reference point product, whether or not it is considered related to the IP or reference point product.

#### 8.1.2 Serious Adverse Events

An SAE is defined as, but not limited to, any untoward medical occurrence that:

- Results in death.
- Is life-threatening.
- Requires inpatient hospitalization or prolongation of existing hospitalization.
- Results in persistent or significant disability/incapacity, or
- Is a congenital anomaly/birth defect.

Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered an SAE when, based on appropriate medical judgment, they may jeopardize the subject or the subject may require medical or surgical intervention to prevent one of the outcomes listed in the above definitions.

Any pre-planned hospitalizations that are known at the time of signing the ICF will not be recorded as SAEs; however, they will be recorded as AEs only. Any AE that occurs during this pre-planned hospitalization will be considered according to the above definitions.


#### 8.2 Assessment of Adverse Events

The Investigator is responsible for obtaining, assessing and documenting all AEs during the study.

#### 8.2.1 Collection of Information

Adverse event information will be collected from the time of signature of the ICF onwards until EOS either by the Investigator via spontaneous reporting or by the use of consistent, open, non-directive questions from study site collaborator (e.g., "Have you had any health problems since the previous visit/How are you feeling since you were last asked?"). At the discretion of the Investigator, the collection of AE information may also be triggered from his/her review of the subject questionnaires and the VAS. However, the main source for AE collection will be the face-to-face interview with the subject.

Information recorded will include: verbatim description of the AE, start and stop dates and times, seriousness, severity (intensity), action taken (e.g. whether or not the AE led to the subject's withdrawal from the study), and outcome (e.g. resolved, withdrawal due to AE).

For each AE the intensity will be graded on a 3-point intensity scale (mild, moderate, severe) using the definitions provided in Section 8.2.3.

Any exacerbation/worsening or increased frequency of an AE or pre-existing condition shall be evaluated and recorded.

Correct medical terminology/concepts are preferred when recording AE terms, and abbreviations must be avoided. Wherever possible, a diagnosis is to be used to describe an AE rather than individual signs and symptoms (e.g. record 'pneumonia' rather than 'fever', 'cough', 'pulmonary infiltrate' or 'septicemia' rather than 'fever' and 'hypotension' following blood sample).

Any AE that meets the serious criteria must be recorded both on the AE report form of the eCRF and on a separate SAE report form (see Section 8.3).

### 8.2.2 Period of Collection

#### 8.2.2.1 Screening Period

All existing health conditions identified during the Screening period will be recorded as concomitant disease and the subject's eligibility for admission to the study will be reviewed. Any AEs which occur during the screening period will be captured by the study site collaborator and assessed by the Investigator in order to establish relationship or relatedness


in respect to study procedures. Only the study procedures-related AEs will be reported in the CSR and in accordance with respective regulatory guidelines.

### 8.2.2.2 Admission Day until the End of Study

From Admission onwards until Day of Discharge, all AEs will be actively collected by the study site collaborator.

Any new, clinically relevant, abnormal finding or worsening of a pre-existing condition/concomitant disease detected during the study will be documented as an AE and/or SAE as described in the safety management plan.

During the safety follow-up period new AEs and/or SAEs will be recorded after spontaneous reporting by the subject. Serious AEs will be reported by the Investigator as described in this document and the Safety Management Plan. Any ongoing AEs/SAEs during the safety follow-up period will be actively followed up by the site until they have been resolved, stabilized (i.e., no worsening of condition), or an acceptable explanation has been found.

At the end of the safety follow-up period all ongoing AEs/SAEs will be followed up by the Investigator on behalf of the Sponsor (see Section 8.3) until they have resolved, stabilized (i.e., no worsening of condition), or an acceptable explanation has been found.

### 8.2.3 Intensity of Adverse Event

For each AE, the intensity will be graded by the Investigator on a 3-point intensity scale (mild, moderate, severe) using the following definitions:

- **Mild**: The AE is easily tolerated and does not interfere with activities of daily living (ADL).
- **Moderate**: The AE interferes with ADL, but the subject is still able to function.
- **Severe**: The AE is incapacitating and requires medical intervention.

# 8.2.4 Relationship to Investigational Product and Relationship to Study Procedures

According to the Council for International Organizations of Medical Sciences VI Working Group, there are no definitive methods for distinguishing most adverse drug reactions (i.e., events that are causally attributed to the IP or reference product) from clinical AEs that occur as background findings in the population and have only temporal association with the IP or reference product.


In general, all AEs and/or SAEs will be assessed by the Investigator as either 'related' or 'not related' to IP or reference product as described below. In addition to the assessment of the relationship of the clinical event to the IP or reference product, the Investigator shall document a potential relationship of the clinical event to any particular study procedure.

- Not related: The temporal relationship of the clinical event to IP administration or a study procedure makes a causal relationship unlikely, or, concomitant medication, therapeutic interventions, or underlying conditions provide a sufficient explanation for the observed event
- **Related**: The temporal relationship of the clinical event to study IP administration or a certain study procedure makes a causal relationship possible, and concomitant medication, therapeutic interventions, or underlying conditions do not provide a sufficient explanation for the observed event.

### 8.2.5 Expectedness

An AE will be regarded as 'unexpected' if its nature or severity is not consistent with information already known about the IP or reference product, and/or has not been previously observed and is not listed in the current IB. The IB provides further detail on signs or symptoms that might be expected with the use of the IP, including information relating to device malfunction or misuse.

NRT gum-related AEs are listed on the product label.

## 8.3 Reporting of Serious Adverse Events

Any SAEs reported or observed during the study after signature of the ICF until the end of the safety follow-up period (i.e. up to 7 days after study Discharge), whether or not attributable to the IP, to any other medication or to any study procedures, or any SAE related to the product and spontaneously reported after the safety follow-up must be reported by the Principal Investigator within 24 hours after first awareness by any party to and to the Sponsor, and the head of the Investigational site.

An SAE report form must be faxed or e-mailed as attachment to:



Philip Morris Products S.A.

Clinical Study Protocol


ZRHR-PK-02-JP

Final 1.0 / 21 June 2013

**Sponsor Contact:** 

**Mobile:** 

E-mail:

Address:

@pmi.com

Philip Morris Products S.A.

R&D Innovation Cube 5 Quai Jeanrenaud 2000 Neuchâtel

Switzerland

The Principal Investigator/the head of the investigational site is responsible for local reporting (e.g., to the IRB) of SAEs that occur during the study, according to local regulations.

Any follow-up information will be detailed in a subsequent SAE report form and sent to and the Sponsor.

The follow-up SAE report form must include the minimum information required for form completion and only changed/new information needs to be specified. Information provided in the follow-up SAE report form supersedes any information that is initially reported.

All SAEs will be followed-up by the Investigator until resolution or until the Investigator considers the event to be stabilized (i.e., no worsening of condition), or an acceptable explanation has been found (e.g., chronic condition).

The SAE report form to be used in this study is provided as a separate document. All SAEs will be recorded on the relevant eCRF page, in addition to the SAE report form.

## 8.4 Reporting of Other Events Critical to Safety Evaluations

### 8.4.1 Abnormal Results of Laboratory Tests

Any clinical safety laboratory test result that is outside of the normal reference range will be reviewed by the Investigator and assessed for clinical relevance. If the Investigator considers the abnormal result to be of clinical relevance, then it must be recorded as a concomitant disease at Screening, or if not present at Screening, as an AE during the study.


The grading scheme shown in (reference to the Common Terminology Criteria for Adverse Events and Common Toxicity Criteria [CTCAE] version 4.03) will be used by the Investigator to assess abnormal laboratory AEs as follows:

- All Grade 1 abnormal laboratory values will be evaluated by the Investigator with respect to baseline value and clinical relevance. If considered to be clinically relevant, the Investigator must report it as an AE. All Grade 2 and higher abnormal laboratory values must be reported as or linked to an AE/concomitant disease.
- If a subject has Grade 2 and higher abnormal laboratory values at Screening, it is at the discretion of the Investigator to enroll the subject or not. This decision must be documented in the source documentation and captured in the eCRF.
- If there is any worsening in grade from Grade 2 and above during the study, the Investigator must report this worsening as an AE.
- Where there is no grading available, the abnormal laboratory value will be evaluated by the Investigator, and assessed for clinical relevance. If considered to be clinically relevant, the Investigator will report it as an AE.
- Any other abnormal clinical laboratory result (including those that are not part of the core safety assessments) can, at the discretion of the Investigator, be reviewed and assessed. Even if they do not meet the criteria of the CTCAE grading scheme (please see above), the Investigator may consider them to be of clinical relevance and, if they are, must report them as AEs.
- In general, laboratory values will be recorded as 'increased <lab parameter>' or 'decreased <lab parameter>' to ensure consistency of recording/coding.

All other information (e.g., relationship to IP, intensity, seriousness, outcome) will be assessed as for other AEs.

### 8.4.2 Abnormal Results of Others Tests or Investigations

An ongoing medical condition or clinically relevant finding detected during the Screening Visit (including elevated laboratory parameters), will be considered a concomitant disease and the subject's eligibility for admission to the study will be reviewed.

Any new, clinically relevant, abnormal finding or worsening of a pre-existing condition detected during the study after Screening until the EOS will be documented as an AE.

Any new onset of symptoms or worsening of pre-existing symptoms identified through the study questionnaires may be documented as AEs at the discretion of the Investigator.

Clinical Study Protocol Final 1.0 / 21 June 2013


### 8.5 Actions and Follow-up

### 8.5.1 Reporting and Follow-up of Pregnancies

For pregnancies detected during the Screening period and prior to first THS 2.2 use, the subject will be considered as a screening failure and removed from the study. No Pregnancy Form will be filled; however, the diagnosed pregnancy must be captured in the Screen Failure eCRF.

All pregnancies occurring after signature of the ICF and diagnosed after first exposure to the IP until completion of the study must be reported by the Investigator.

Any pregnancy potentially associated to exposure to the IP, including pregnancies spontaneously reported to the Investigator after the EOS must be reported by the Investigator and followed-up. Potential association with exposure to the IP is defined as the conception date being calculated before the last exposure to the IP.

The Investigator will complete a Pregnancy Form (provided as a separate document) for all pregnancies diagnosed (including positive urine pregnancy tests).

The procedure to report a pregnancy and provide any additional/follow-up information to and the Sponsor must be followed in the same manner and within the same timelines as described for an SAE (see Section 8.3). In addition, each pregnancy has to be reported as a non-serious AE. No invasive procedures, including drawing of blood, must be done in such subjects after the discovery of pregnancy.

United BioSource Corporation Safety will follow-up pregnancies only if they were detected after first product use (i.e., after THS 2.2 test on Admission Day). If pregnancies are to be followed-up, they will be followed-up until an outcome is reached (e.g., normal delivery, spontaneous abortion, or voluntary termination). Any pregnancy complications, adverse pregnancy outcomes, or maternal complications will be recorded.

The Principal Investigator/head of the investigational site is responsible for informing the IRB of any pregnancy that occurs during the study and its outcome, according to local regulations.

### 8.5.2 Adverse Events Leading to Withdrawal

Subjects who are withdrawn from the study because of an AE will undergo the procedures, as described for the Day of Discharge, as soon as possible and will enter the period of safety follow-up. The Investigator will follow-up these AEs until they have resolved, stabilized (i.e., no worsening of condition), or an acceptable explanation has been found.

Clinical Study Protocol Final 1.0 / 21 June 2013 

### 8.5.3 Investigational Device Misuse

Any occurrences of the THS Tobacco Stick Holder or THS Charger misuse (use not in accordance with its label and instruction) by a subject, will be documented by the Investigator or his/her designated staff using a Device Issue Log.

Investigational device misuse may result in use-related hazards.

Use-related hazards are derived from the US Food and Drug Administration Medical Device Use-Safety Guidance (FDA, 2012b):

- Hazards caused specifically by how a device is used.
- Unanticipated use scenarios (e.g., modification of Charger, applying any chemicals, using CCs, mechanical damage of the unit, etc.) that result in hazards must be documented and reported by the Investigator.

According to FDA Medical Device Regulation, data should be collected regarding the use related hazards that have occurred with the device and when information pertaining to device use safety is extensive, it is helpful to provide it in summary form that highlights the most important issues, considerations, resolutions, and conclusions. The level of detail of device use documentation submitted should be consistent with the level of concern of use-related hazards for the device.

Furthermore, any misuse of the THS Tobacco Stick Holder or THS Charger, that lead to an AE/SAE will follow the same processes as described above.

### 8.5.4 Investigational Device Malfunction

Any occurrences of malfunction of the Tobacco Stick Holder or Charger will be documented by the Investigator or his/her designated study collaborator using a Device Issue Log.

Furthermore, any malfunctions of the Tobacco Stick Holder or Charger that lead to an AE/SAE will follow the same processes as described above.


#### 9 STUDY ACTIVITIES

A detailed schedule of assessments can be found in Appendix 1. The time points shown are to be considered the time of assessment for the first subject. As not all subjects can be treated at the same time, a short time window will be implemented for subsequent subjects. Measurements not conducted at the exact time point, but conducted within the given time window (if applicable) do not constitute a protocol deviation but an accepted variability for the given time point.

In general, if no start time for the procedure is provided, then the procedure can be performed at any time during the day.

### 9.1 Screening Visit

The Screening Visit will be performed within 4 weeks (Day -29 to Day -2) prior to Admission (Day -1). Subjects will attend the investigational site in at least a 10-hour fasting state for clinical laboratory to be assessed.

The following assessments will be performed at the Screening Visit (Table 4) (the sequence of the assessment will be at the discretion of the site but all of them must be done after signature of the ICF).

Table 4 Time Schedule – Screening Visit

| Time | Blood sample | Procedures | Additional information |
|---|---|---|---|
| Start of procedure | | | |
| | | Informed consent/Subject Information Sheet | |
| | | Demographic data | On the day of ICF signature |
| | | Advice on the risks of smoking and debriefing | |
| | | Smoking history | |
| | | Willingness to abstain from smoking in the next 3 months | |
| | | Readiness to accept interruptions of smoking for up to 4 days | |
| | | FTND questionnaire | |
| | | Prior/concomitant medication | |


| ====================================== | 1 11141 1.0 / 21 0 4110 2010 | 1 480 75 01 122 |
|---|---|---|
| | Medical history/concomitant diseases | |
| | Vital signs (pulse rate, systolic and diastolic blood pressure, respiratory rate) | At least 5 min in supine position prior to measurement |
| | Height, weight, including calculated BMI | |
| V | Clinical laboratory parameters (hematology, urine analysis, clinical chemistry) | At least in 10 hours fasting condition |
| V | Serology for HIV and Hepatitis B and C | |
| | Identification of current CC brand | |
| | Urine drug screen | |
| | Alcohol breath test | |
| | Urine pregnancy test for female subjects | |
| | THS 2.2 and NRT gum product demonstration | |
| | Spirometry without short-acting bronchodilator first, and then with | Has to be done at least 1 hour after smoking |
| | ECG | At least 10 min in supine position prior to recording |
| | AE/SAE questioning | If the Screening Visit is<br>performed on two separate days<br>the AE/SAE questions will be<br>asked again |
| | Physical examination | |
| | Chest X-ray (if not performed 6 months prior to Screening) | |
| | Urine cotinine screening test | |
| | T 1 ' / 1 ' ' ' | |

Clinical Study Protocol

Final 1.0 / 21 June 2013

Abbreviations: AE = Adverse event; BMI = Body mass index; CC = Conventional cigarette(s); ECG = Electrocardiogram; FTND = Fagerström Test for Nicotine Dependence (revised version); HIV = Human immunodeficiency virus; ICF = Informed consent form; NRT gum = Nicotine replacement therapy gum; SAE = Serious adverse event; THS 2.2 = Tobacco Heating System 2.2

Inclusion/exclusion criteria

# 9.2 Admission

Philip Morris Products S.A.

ZRHR-PK-02-JP

The following assessments will be performed at Admission (Day -1) (Table 5):

Clinical Study Protocol


ZRHR-PK-02-JP

Final 1.0 / 21 June 2013


Table 5. Time Schedule – Day -1 Admission

| Time | Blood<br>sample | Procedures | Additional information |
|---|---|---|---|
| Start of procedure | | | |
| | | AE/SAE recording, concomitant medication | All day |
| | | Advice on the risks of smoking and debriefing | |
| | | Readiness to accept interruptions of smoking for up to 4 days | |
| | $\sqrt{}$ | trans-3'-hydroxycotinine and cotinine (CYP2A6 activity) in plasma | The subject should not have smoked in the morning until this assessment |
| | | | Must be done prior to smoking |
| | | Spirometry | Must be done prior to smoking |
| 6:30 AM | | Beginning of smoking period | |
| | $\sqrt{}$ | Clinical laboratory parameters (hematology, urine analysis, clinical chemistry) | To be done at least in 10-hour fasting condition |
| Prior to 10:00 AM | | Breakfast | |
| Prior to 11:30 AM | | Urine pregnancy test for all female subjects | |
| Prior to 11:30 AM | | Urine cotinine screening test | |
| Prior to 11:30 AM | | Urine drug screen | |
| Prior to 11:30 AM | | Vital signs | At least 5 min in supine position prior to measurement |
| Prior to 11:30 AM | | Physical examination, weight and calculated BMI | |
| Prior to 11:30 AM | | Identification of current CC brand | |

| Philip Morris Products S.A. | Clinical Study Protocol | Confidential |
|---|---|---|
| ZRHR-PK-02-JP | Final 1.0 / 21 June 2013 | |
| Prior to 11:30 AM | Smoking history | |
| Prior to 11:30 AM | Alcohol breath test | |
| Prior to 11:30 AM | CO breath test | |
| Prior to 2:30 PM | Lunch | |
| Afternoon | Snacks | |
| | Product test for THS 2.2 and NRT gum | The THS 2.2 test should be done first and then the NRT gum test. |
| | | Subject on NRT gum should chew slowly for $35 \pm 5$ minutes, while spacing between each chew |
| | Inclusion/exclusion criteria | |
| | Enrolment | |
| Prior to 9:00 PM | Dinner | |
| 11:00 PM | End of smoking period | |

Abbreviations: AE = Adverse event; BMI = Body mass index; CC = Conventional cigarette(s); CO = Carbon monoxide; CYP2A6 = Cytochrome P450 2A6; NRT gum = Nicotine replacement therapy gum; SAE = Serious adverse event; THS 2.2 = Tobacco Heating System 2.2.

# 9.3 Investigational Period

# 9.3.1 Days of Smoking Abstinence (Day 0 and Day 2)

On the days of SA (Day 0 and Day 2) the following assessments will be performed (Table 6 and Table 7):

Table 6. Time Schedule – Day 0 Washout

| Time | Blood<br>sample | Procedures | Additional information |
|---|---|---|---|
| Start of procedure | | | |
| | | Nicotine abstinence | All day |

| Philip Morris Products S.A. | Clinical Study Protocol | Confidential |
|---|---|---|
| ZRHR-PK-02-JP | Final 1.0 / 21 June 2013 | |
| | Support during nicotine abstinence as required | All day |
| | AE/SAE recording, concomitant medication | All day |
| | Randomization | At any time of the day |
| 06:30AM-09:00 AM | Assessment of cough | |
| Prior to 10:00 AM | Breakfast | |
| 8:00 AM-9:30 AM | CO breath test | |
| 10:00 AM-11:30 AM | Vital signs | At least 5 min in supine position prior to measurement |
| 12:00 PM-1:30 PM | CO breath test | |
| Prior to 2:30 PM | Lunch | |
| 4:00 PM-5:30 PM | CO breath test | |
| Afternoon | Snacks | |
| Prior to 9:00 PM | Dinner | |
| 8:00 PM-9:30 PM | CO breath test | |

Abbreviations: AE = Adverse event; CO = Carbon monoxide; SAE = Serious adverse event.


Table 7. Time Schedule - Day 2 Washout

| Time | Blood<br>sample | Procedures | Additional information |
|---|---|---|---|
| Start of procedure | | | |
| | | Nicotine abstinence | All day |
| | | Support during nicotine abstinence as required | All day |
| | | AE/SAE recording, concomitant medication | All day |
| | $\sqrt{}$ | Plasma nicotine PK sample | 24 hrs +5 min after $T_0$ of Day 1 $(T_{15})$ |
| | | Assessment of cough | 24 hrs minus 5 min after $T_0$ of Day 1 |
| Prior to 10:00 AM | | Breakfast | |
| 8:00 AM-9:30 AM | | CO breath test | |
| 10:00 AM-11:30 AM | | | At least 5 min in supine position prior to measurement |
| 12:00 PM-1:30 PM | | CO breath test | |
| Prior to 2:30 PM | | Lunch | |
| 4:00 PM-5:30 PM | | CO breath test | |
| Afternoon | | Snacks | |
| Prior to 9:00 PM | | Dinner | |
| 8:00 PM-9:30 PM | | CO breath test | |

Abbreviations: CO = Carbon monoxide; PK = Pharmacokinetic; T = Time point.

Clinical Study Protocol Final 1.0 / 21 June 2013 Confidential


# 9.3.2 Days of Single Use (Day 1 and Day 3)

On the days of single use (Day 1 and Day 3) the following assessments will be performed (Table 8):

Clinical Study Protocol Final 1.0 / 21 June 2013 Confidential


Table 8. Time Schedule - Day 1 and Day 3 Product Use

| Time | Blood<br>sample | Procedures | Additional information |
|---|---|---|---|
| Start of procedure | | | |
| | | Optional: light snacks<br>prior to first blood draw<br>of the day | |
| | | AE/SAE recording, concomitant medication | All day |
| | | Craving questionnaire (QSU-brief) | For subjects on THS 2.2 or on CC: First sample within 15 min prior to $T_0$ , 9 assessments thereafter in relation to $T_0$ : 15 min, 30 min, 45 min, 60 min, 2 hr, 4 hrs, 6 hrs, 9 hrs, and 12 hrs after $T_0$ , with an allowed time window of +10 min each |
| | | | For subjects on NRT gum: First sample within 15 min prior to $T_0$ , 9 assessments thereafter in relation to $T_0$ : 20 min, 30 min, 45 min, 60 min, 2 hr, 4 hr, 6 hrs, 9 hrs, and 12 hrs after $T_0$ , with an allowed time window of +10 min each |

| Philip Morris Products S.A. | Clinical Study Protocol | Confidential |
|-----------------------------|--------------------------|----------------|
| ZRHR-PK-02-JP | Final 1.0 / 21 June 2013 | |

| | Plasma nicotine sample | For subjects on THS 2.2 or on CC: a total of 16 blood samples will be taken for a 24-hour profile (Day 1 and Day 3). The first blood sample will be taken within 15 min prior to T <sub>0</sub> and 15 samples thereafter in relation to T <sub>0</sub> : T <sub>1</sub> after 2 min +1 min, T <sub>2</sub> after 4 min +1 min, T <sub>3</sub> after 6 min +1 min, T <sub>4</sub> after 8 min +1 min, T <sub>5</sub> after 10 min +1 min, T <sub>6</sub> after 15 min +2 min, T <sub>7</sub> after 30 min +2 min, T <sub>8</sub> after 45 min +2 min, T <sub>9</sub> after 60 min +3 min, T <sub>10</sub> after 2 hrs +5 min, T <sub>11</sub> after 4 hrs +5 min, T <sub>12</sub> after 6 hrs +5 min, T <sub>13</sub> after 9 hrs +5 min, T <sub>14</sub> after 12 hrs +5 min, and T <sub>15</sub> after 24 hrs +5 min (this sample will be drawn during the day following product use, i.e., wash-out). For subjects on NRT gum: A total of 16 blood samples will be taken for a 24-hour profile (Day 1 and Day 3). The first blood sample will be taken within 15 min prior to T <sub>0</sub> and 15 samples thereafter in relation to T <sub>0</sub> : T <sub>1</sub> after 10 min + 1 min, T <sub>2</sub> after 20 min + 1 min, T <sub>3</sub> after 25 min + 1 min, T <sub>4</sub> after 30 min + 1 min, T <sub>5</sub> after 35 min + 1 min, T <sub>6</sub> after 40 min + 1 min, T <sub>7</sub> after 45 min + 1 min, T <sub>8</sub> after 60 min + 3 min, T <sub>9</sub> after 2 hrs + 5 min, T <sub>10</sub> after 3 hrs + 5 min, T <sub>11</sub> after 4 hrs + 5 min, T <sub>12</sub> after 6 hrs + 5 min, T <sub>13</sub> after 9 hrs + 5 min, T <sub>14</sub> after 12 hrs + 5 min, and T <sub>15</sub> after 24 hrs +5 min (this sample will be drawn during the day following product use, i.e., wash-out). |
|---|---|---|
| $\sqrt{}$ | COHb blood sampling | Five blood samples to be taken, first sample within 15 min prior to T <sub>0</sub> , then after 15 min +2 min, 60 min +3 min, 4 hrs +5 min, 12 hrs +5 min |
| | CO breath test | First test to be done within 15 min prior to $T_0$ |
| | Assessment of cough | Has to be done prior to product use |

Confidentiality statement: Data and information contained in this document are considered to constitute trade secrets and confidential commercial information, and the legal protections provided to such trade secrets and confidential information are hereby claimed under the provisions of applicable law. No part of this document may be publicly disclosed without the written consent of Philip Morris Products S.A.

Start of single product use

6:00 AM-9:00 AM

| Philip Morris Products S.A. | Clinical Study Pro | tocol Confidential |
|---|---|---|
| ZRHR-PK-02-JP | Final 1.0 / 21 June | 2013 |
| Prior to 10:00 AM | Breakfast | |
| 10:00 AM-11:30 AM | Vital signs | At least 5 min in supine position prior to measurement |
| 10:00 AM-11:30 AM | ECG | At least 10 min in supine position prior to recording |
| 12:00 PM-1:30 PM | CO breath test | |
| Prior to 2:30 PM | Lunch | |
| 4:00 PM-5:30 PM | CO breath test | |
| Afternoon | Snacks | |
| Prior to 9:00 PM | Dinner | |
| 8:00 PM-9:30 PM | CO breath test | |
| 8:00 PM-11:00 PM | Product evaluation<br>questionnaire (MCEQ;<br>only in sequence 1 and 2) | |
| | Collection of used<br>Tobacco Sticks and CC<br>butts and NRT gum | After the product use |

Abbreviations: AE = Adverse event; CC = Conventional cigarette(s); CO = Carbon monoxide; COHb = Carboxyhemoglobin; ECG = Electrocardiogram; MCEQ = Modified Cigarette Evaluation Questionnaire; NRT gum = Nicotine replacement therapy gum; QSU-brief = Questionnaire of Smoking Urges brief; SAE = Serious adverse event; T = Time point; THS 2.2 = Tobacco Heating System 2.2

# 9.4 Day of Discharge

The following assessments will be conducted prior to the time of Discharge on Day 4 (or after a subject is prematurely withdrawn from the study) (Table 9):

ZRHR-PK-02-JP

Clinical Study Protocol Final 1.0 / 21 June 2013 

Table 9. Time Schedule – Day 4 Discharge

| Time | Blood sample | Procedures | Additional information |
|---|---|---|---|
| Start of procedure | | | |
| | | AE/SAE recording, concomitant medication | All day |
| | V | Plasma nicotine: PK sample | 24 hrs +5 min since T <sub>0</sub> of Day 3 (T <sub>15</sub> ) |
| | | Assessment of cough | 24 hrs minus 5 min since $T_0$ of Day 3 |
| | $\checkmark$ | Clinical laboratory parameters (hematology, urine analysis, clinical chemistry) | Has to be done in at least 10-hour fasting condition |
| | | Spirometry | Has to be done prior to smoking |
| Prior to 10:00 AM | | Breakfast | |
| Prior to discharge | | CO breath test | |
| Prior to discharge | | Urine pregnancy test in all female | |
| Prior to discharge | | Vital signs | At least 5 min in supine position prior to measurement |
| Prior to discharge | | Physical examination, weight and calculated BMI | |
| Prior to discharge | | Advice on the risks of smoking and debriefing | |
| | | Time of discharge | |

Abbreviations: AE = Adverse event; BMI = Body mass index; CO = Carbon monoxide; PK = Pharmacokinetic; SAE = Serious adverse event; T = Time point.

Smoking will be allowed after spirometry has been conducted.

Clinical Study Protocol Final 1.0 / 21 June 2013 Confidential


# 9.5 Safety Follow-up Period

All subjects participating in the product trial on Day -1 and are not enrolled into the study will enter a 7-day safety follow-up period.

After the time of Discharge at Day 4 (or if prematurely withdrawn from the study), subjects will enter a 7-day safety follow-up period.

During the 7-day safety follow-up period, there will be spontaneous reporting by the subject of new AEs and new SAEs. Any ongoing AEs/SAEs will be actively followed up by the site.

Any AEs or SAEs that are ongoing at the end of the 7-day safety follow-up period will be handled as described in Section 8

# 9.6 Early Termination Procedures

The Day of Discharge assessments will be performed as early termination procedures (see Section 9.4). Early termination procedures will be the same as those described in the Day of Discharge.


## 10 QUALITY CONTROL AND QUALITY ASSURANCE

# 10.1 Monitoring

The Clinical Research Associate (CRA) ("Monitor") will be responsible for the monitoring of the study. Monitoring will be performed according to CRO's SOPs and as per the agreed monitoring plan with the Sponsor.

The Principal Investigator/head of the investigational site shall permit the Monitor to review study data as frequently as considered necessary to ensure that data are being recorded in an adequate manner and that protocol adherence is satisfactory.

The Investigator shall access medical records for the Monitor in order that entries in the eCRFs may be verified. The Investigator, as part of their responsibilities, is expected to ensure that the study adheres to GCP requirements.

An Investigator's meeting will be held prior to the site initiation visit. During this meeting, the general training of the study procedures and specific training on selected procedures will be done and documented.

Subsequent to the Investigator's meeting, and before the first subject is screened into the study, site initiation visit will be conducted by the Monitor and, if necessary, with Sponsor or its authorized representative. The purpose of the site initiation visit will be detailed in the monitoring plan.

Communication by telephone, mail, and e-mail may be used as needed to supplement site visits. The Investigator and study personnel will cooperate with the Monitor, provide all appropriate documentation, and will be available to discuss the study.

The Monitor and the Sponsor's personnel will be available between visits, should the Investigator or other study collaborators at the sites need information and advice.

Site visits will be made at regular intervals during the study. The frequency of the monitoring visits will be defined in the monitoring plan agreed with the Sponsor.

The Investigator, or a designated member of the Investigator's study collaborators, must be available during the monitoring visit to review the data and resolve any queries, and to allow direct access to the subject's records for source data verification.


# 10.2 Training of Study Collaborator

A formal meeting (Investigator's meeting) will be conducted prior to site initiation. During this meeting, the Sponsor or its authorized representative will discuss the requirements of the clinical study protocol and related documents and will also provide training in the relevant systems and other study-specific procedures. The activities of the Investigator's meeting will be described in the monitoring plan.

In addition to the Investigator meeting, the Investigator will ensure that appropriate training relevant to the study is provided to all study collaborator involved in the study, and that any new information relevant to the performance of this study is forwarded to the study collaborator involved in a timely manner. The record of all individuals involved in the study will be maintained in the Site Investigator File.

# 10.3 Audits and Inspections

Good Clinical Practice regulations require that there are independent inspections of clinical program activities. Such inspections may be performed at any time before, during and/or after the study.

Authorized representatives of the Sponsor, regulatory agencies and/or an IRB may perform audits or inspections, including source data verification. The purpose of an audit or inspection is to systematically and independently examine all study-related activities and documents to determine whether these activities were conducted, and data were recorded, analyzed, and accurately reported according to the protocol, ICH/GCP guidelines, and any applicable regulatory requirements. The Principal Investigator/head of investigational site will contact the Sponsor or the authorized representative immediately, if contacted by a regulatory agency about an inspection at their site.

The Investigator and study collaborator are responsible for maintaining a comprehensive and accurate filing system of all study-related documentation that will be suitable for inspection at any time by the Sponsor, its authorized representative, and/or regulatory agencies. In signing this protocol, the Investigator understands and agrees to provide access to the necessary documentation and files.


### 11 DATA MANAGEMENT ACTIVITIES

All Data Management Activities will be described in detail in the Data Management Plan (DMP) and documents specified therein.

# 11.1 Data Capture

# 11.1.1 Case Report Forms and Study Records

With the exception of the subject reported outcome data, all results from the clinical assessments will be recorded in the Source Documents by the Investigator and then captured in the eCRFs at the study site. The subject questionnaires and the VAS will be entered by the subject directly in the ePRO device. Trained study personnel will be responsible for capturing the data from the observations, tests, and assessments specified in the protocol in the Source Documents and then transferring the data into the eCRF according to the eCRF Completion Guidelines.

The Principal Investigator has ultimate responsibility for the collection and reporting of all data related to the clinical study and ensuring that the data are accurate, authentic/original, legible, timely (contemporaneous), enduring, and available when required. The eCRF must be signed by the Investigator to attest that the data contained in the eCRF are true and accurate. Any corrections made to Source Documents must be clearly recorded, without obscuring the original values and be accompanied by the date of change, reason for change, and identification of the person making the change. The eCRF for each subject will be checked against the Source Documents at the study site by the CRA. Instances of missing or unclear data will be discussed with the Investigator for resolution. An eCRF will be generated for all subjects that sign the informed consent.

### 11.1.2 Protocol Deviations

All protocol deviations will be entered into the Clinical Trial Management System (CTMS) or other approved format.

Information from the Source Documents will represent the primary source of protocol deviations. Information following site monitoring and other manual reviews will be documented in the site visit reports, follow-up letters, audit documentation, or other manual review and will be recorded and tracked in the CTMS or other approved format. Telecommunications and other verbal communications regarding deviations will be considered and handled as important communication, documented and tracked as protocol deviations, as necessary.

Philip Morris Products S.A.

Clinical Study Protocol


ZRHR-PK-02-JP

Final 1.0 / 21 June 2013


Individual entries for protocol deviations that are recorded in the CTMS, or other approved format, following site monitoring and other manual reviews will be reviewed against the individual data points in the eCRF database but will not be formally reconciled with the eCRF database (e.g., their description or occurrence date). The overall procedure for managing protocol deviations are described in the SOPs of the CRO Data Management Team. All deviations will be reviewed periodically, as determined at study start, to identify trends to improve monitoring and/or potential impact on the statistical analysis.

# 11.2 Data Handling

All study data will be managed by the Data Management Team at the CRO. The overall procedures for quality assurance of clinical study data are described in the SOPs of the CRO Data Management Team. The Data Management Team at CRO will prepare a DMP, to be reviewed and approved by the Sponsor, prior to the start of the study. This document will describe, in detail, the Data Management related procedures and processes.

All data of all subjects enrolled and screening failures who experience an AE during the study (from time of informed consent to end of the safety follow-up period) will be captured and stored in the study database.

All data collected during the study is property of the Sponsor irrespective of the location of the database and the Data Management CRO.

#### 11.2.1 Data Validation

The data will be validated as defined in the DMP and Data Validation Specifications. Discrepancies will be reported as defined in DMP and Data Validation Plan.

Data queries will be raised for discrepant or missing data. All changes to data will be captured in the database with a comprehensive audit trail.

### 11.2.2 Coding

Adverse events, medical/surgical history, and prior/concomitant medication will be classified according to the terminology of the latest version of the following Dictionaries, at time of coding the first entry:

Medical history: Medical Dictionary for Regulatory Activities (MedDRA®)

Adverse events: MedDRA®

Medications: WHO Drug Dictionary Enhanced and Anatomical Therapeutic

and Chemical classification system

Clinical Study Protocol Final 1.0 / 21 June 2013


THS 2.2 device issues C54451/Medical\_Device\_Problem\_Codes\_FDA\_CDRH and/or malfunctions:

#### 11.2.3 Database Lock

When all outstanding Data Management issues have been resolved and all validation, quality review, and cleaning activities are complete, the database or selected data is/are declared soft locked. Access to change data in the soft-locked database or to change selected data at this time is limited

After the data is reviewed by the Sponsor, resolution of all raised queries and QC of the changed data, database, or selected data upon Sponsor approval as applicable, is declared locked.

Any changes to the database after that time can only be made by written agreement between the Sponsor and the Data Management and Statistical Team at the CRO. Any of those changes must be documented in the database log file.

After study completion, the study database will be transferred to the Sponsor in the format specified in the DMP in Clinical Data Interchange Standards Consortium's Study Data Tabulation Model Data Structure Specifications.


### 12 PLANNED STATISTICAL METHODS

### 12.1 General Considerations

An incomplete block design will be adopted in this study with every subject being exposed to 2 out of the 3 study products (CC, THS 2.2, and NRT gum) to allow comparisons between THS 2.2 and CC in Group-1 (sequence 1 and 2), and between THS 2.2 and NRT gum in Group-2 (sequence 3 and 4).

Full details of the statistical analysis will be given in a SAP. Any changes to the planned statistical methods will be documented in the Clinical Study Report. The statistical evaluation will be performed using SAS®, version 9.2 or later.

### 12.1.1 Stratification Criteria

For analysis, the following stratification criteria will be used:

- Sex (male and female)
- CC nicotine level at Admission (ISO nicotine levels ≤0.6 mg and 0.6 to 1 mg)

In addition, for the safety data, the analysis will be stratified by sequence and by study periods (Screening, product test, product exposure, and safety follow-up period).

# 12.1.2 Definitions for Statistical Data Analysis

Unless otherwise stated, for the purposes of statistical analyses, baseline is defined as the last available time point prior to T<sub>0</sub> on Day 1, from 6:00 AM to 9:00 AM.

### 12.1.3 Descriptive Statistics

All data will be presented in listings, ordered by sequence and subject, unless otherwise specified.

Descriptive statistics for continuous variables (number of subjects [n], number and percentage of subjects with missing data, mean, standard deviation, median, first and third quartiles, minimum and maximum for continuous data, and the n and absolute and relative [%] frequency for categorical data) will presented by exposure and overall at each time point, where applicable.

Descriptive statistics for PK parameters will also include the geometric mean and coefficient of variation (CV).


Baseline, admission and screening data (i.e., anything prior to product exposure) will be summarized by sequence and overall where appropriate

## 12.1.4 Handling of Missing Values and of Values outside the Detection Limits

In general, missing data will not be imputed in this study, due to the nature of the measurements and the short periods of exposure and use. However, for questionnaire data total scores and domain or subscale scores may use a certain degree of imputation by averaging across individual item scores. Further details will be provided in the SAP.

Values below the lower limit of quantification (LLOQ) will be imputed using 0.5 x LLOQ. For values above the upper limit of quantification (ULOQ), i.e., preceded by a ">", for example ">xx", the numerical xx will be used for calculation and reporting in summary tables. The number of values below LLOQ or above ULOQ will be presented in each summary table.

# 12.1.5 Significance Level for Inferential Analysis

For all endpoints, unless otherwise stated, statistical tests will be two-sided and conducted at the 5% significance level and all quoted confidence intervals will be two-sided 95% CIs.

No formal adjustment of the test-wise alpha level for multiple testing is necessary, as no claim will be made based on the outcome of the individual tests.

# 12.2 Determination of Sample Size and Power Consideration

A total of 62 subjects will be randomized. This sample size is the sum of the sample size requirements for the THS 2.2:CC comparison and the THS 2.2:NRT gum comparison (as described in detail below).

The estimates for the within-subject CV for nicotine  $C_{max}$  (36%) and  $AUC_{(0-last)}$  (21%) are based on the data collected in the ZRHX-PK-02 clinical study (ZRHX-PK-02, 2012) comparing the nicotine PK profiles of Tobacco Heating System 2.1, the predecessor of THS 2.2 (regular tobacco stick) and CC. In the absence of data comparing THS and NRT gum, the same CVs were assumed for the calculation of the sample size related to the THS 2.2:NRT gum comparison.

Anticipated mean  $C_{max}$  and  $AUC_{(0-last)}$  for THS 2.2 and CC were based on data from the ZRHX-PK-02 study (ZRHX-PK-02, 2012). Anticipated mean  $C_{max}$  and  $AUC_{(0-last)}$  for NRT gum were based on data reported by Dautzenberg et al., 2007.

The sample sizes of this study assume a drop-out rate no larger than 10%.


ZRHR-PK-02-JP

Final 1.0 / 21 June 2013


Sample size calculations were conducted using SAS<sup>®</sup> version 9.2 for the 95% CI of the mean differences between paired observations (proc power onesamplemeans) in the natural log scale (Senn, 2002). The SAS<sup>®</sup> implementation of the method published by Beal, 1989 was adopted to estimate the probability of obtaining at most the target 95% CI of  $\pm 20\%$ .

### THS 2.2:CC comparison

A total of 44 subjects are needed to estimate the mean  $C_{max}$  parameter ratio between THS 2.2 and CC with a 90% probability of obtaining a margin of error (95% CI) of at most  $\pm 20\%$ , assuming that THS 2.2 have a nicotine  $C_{max}$  similar to CC (ratio equal to 1.00). This sample size is sufficient to provide 90% probability of obtaining a margin of error of at most  $\pm 20\%$  for the AUC<sub>(0-last)</sub> ratio between THS 2.2 and CC, assuming a similar extent of nicotine absorption for the 2 products (ratio equal to 1.00).

# THS 2.2:NRT gum comparison

A total of 18 subjects are needed to estimate the mean  $AUC_{(0\text{-last})}$  parameter ratio between THS 2.2 and NRT gum with a precision allowing for the lower bound of the 95% CI exceeding 1.00, with 90% power, assuming a geometrical ratio between THS 2.2 and NRT gum of 1.28. This sample size is sufficient to provide 90% power of obtaining a lower bound of the 95% CI of  $C_{max}$  ratio between THS 2.2 and NRT gum, exceeding 1.00, assuming a geometrical mean ratio between THS 2.2 and NRT gum of 2.00.

# 12.3 Analysis Populations

All analyses will be based on actual product exposure. All endpoints (other than safety) will be analyzed using the PK analysis sets. Safety will be analyzed using the safety population.

# 12.3.1 PK Populations

The analysis populations for the PK endpoints are composed of two analysis sets to allow the comparison between THS 2.2 and NRT gum separately from the comparison between THS 2.2 and CC.

The PK populations consist of all the randomized subjects who give informed consent, completed at least one of the single use Day 1 or Day 3, and for whom at least one PK parameter can been derived. Only subjects without major protocol deviations (to be defined in the SAP) will be included in the PK analysis sets.

# 12.3.2 Safety Population

The safety population consists of all the subjects who give informed consent and have at least one exposure to THS 2.2 (including the product test at Admission Day).


# 12.4 Demographics and Baseline Characteristics

Demographic and other baseline characteristics will be reported for the PK and safety populations. Appropriate summary statistics will be provided as described in Section 12.1.3.

# 12.5 Primary Endpoints

# 12.5.1 Primary Endpoint Analysis Variables

Nicotine PK parameters will be derived from plasma nicotine versus time data using a non-compartmental technique. In particular:

 $C_{max}$  Maximum observed plasma concentration.  $C_{max}$  will be reported as long as there is at least one quantifiable concentration post-exposure

AUC<sub>(0-last)</sub> Area under the plasma concentration-time curve from start of product use to the time of the last quantifiable concentration (linear trapezoidal method).

# 12.5.2 Baseline Comparability

Not applicable.

# 12.5.3 Descriptive Analysis

Primary endpoints will be summarized as described in Section 12.1.3.

An analysis of variance (ANOVA) will be conducted on  $AUC_{(0-last)}$  and  $C_{max}$  endpoints in the natural logarithmic scale. The model will include terms for sequence, subjects within sequence, period and product exposure as fixed effect factors. The results of this analysis for each of  $AUC_{(0-last)}$  and  $C_{max}$  are presented in terms of adjusted geometric least square means and 95% CIs for the THS 2.2 :CC and THS 2.2:NRT gum ratios.

This approach is consistent with the guidelines in the European Medicines Agency's guidelines for bioequivalence investigations (EMA, 2008) and FDA's Center for Drug Evaluation and Research (FDA, 2001). Carry-over effect will not be tested, as it cannot be statistically distinguished from the interaction between treatment and period in a 2x2 crossover design (ICH E9, 1998).

A sensitivity analysis will be conducted should there be 20% or more missing PK parameter values, by repeating the above analyses using mixed effects ANOVA model in the natural log scale, with a restricted maximum likelihood method to estimate mean differences and

Clinical Study Protocol Final 1.0 / 21 June 2013 Confidential


variances as suggested by FDA (FDA, 2001). Subjects within sequence will be used as random effects and fixed effects are period, sequence, and product exposure. To evaluate the sensitivity to the distributional assumptions, point and interval estimates will also be estimated by means of the percentile bootstrap technique, using 2000 bootstrap samples which preserve the number of subjects per sequence.

# 12.5.4 Confirmatory Analyses

Given that the objective of this study is to determine the point estimate and precision of the ratio of THS 2.2:CC for  $C_{max}$  and  $AUC_{(0-last)}$ , there is no statistical hypothesis to be tested.

# 12.6 Secondary Endpoints

# 12.6.1 Secondary Endpoint Analysis Variables

Nicotine PK parameters will be derived as follows:

 $t_{max}$  Time of maximum observed plasma concentration.  $t_{max}$  will be reported as long as there is at least one quantifiable concentration post-exposure

AUC<sub>(0-t')</sub> Area under the plasma concentration-time curve from start of product use to the subject-specific time of maximum nicotine concentration following CC or NRT gum (linear trapezoidal method)

AUC $_{(0-\infty)}$  Area under the plasma concentration-time curve from start of product use extrapolated to infinite time, according to:

$$AUC_{0-\infty} = AUC_{0-last} + \left(\frac{C_{last}}{\lambda z}\right)$$

Where  $C_{last}$  is the last quantifiable concentration and  $\lambda_z$  is the terminal elimination rate constant

 $\lambda_z$  Terminal elimination rate constant, estimated by linear regression analysis of the natural log-transformed concentration-time data

 $t_{1/2}$  Terminal elimination half-life, derived as  $ln(2)/\lambda_z$ 

More details on PK parameter derivations will be provided in the SAP.


Subjective effects of using THS 2.2 as compared to CC and NRT gum will be evaluated by analyzing domain scores of the QSU-brief and MCEQ. Full details of questionnaire domain scores derivation will be provided in the SAP.

## 12.6.2 Baseline Comparability

Not applicable.

# 12.6.3 Descriptive Analysis

In general, secondary endpoints will be summarized using the approach described in Section 12.1.3.

The following analyses will be conducted in both Group-1 and Group-2 PK analysis sets:

- The AUC<sub>(0- $\infty$ )</sub>, AUC<sub>(0-t')</sub>, and t<sub>1/2</sub> will be analyzed using the same approach adopted for the primary endpoints. No statistical analysis will be performed on the elimination rate constant  $\lambda_z$ . Data will be summarized and presented together with 95% CI.
- The Hodges-Lehmann 95% CI estimates for the median t<sub>max</sub> differences will be presented (Lingling, 2008).
- The use of random effects model is suggested in the context of the analysis of subjective effects of smoking (Shiffman et al., 2004). Mixed effects ANOVA with the same model terms as planned for the sensitivity analysis of the primary endpoints will be adopted for the analysis of QSU-brief, including all of the different assessment time points as repeated measurements. The analysis will not be adjusted for the assessment prior to T<sub>0</sub> (Fleiss et al, 1985).
- Levels of exhaled CO and of blood COHb will be summarized by means of descriptive statistics reported by exposure. Analysis of COHb levels will be conducted using a mixed model for repeated measures, the same approach as for the QSU-brief.

The following analyses will be conducted only in Group-1 PK analysis set:

 Mixed effects ANOVA with the same model terms as planned for the sensitivity analysis of the primary endpoints will be adopted for the analysis of the MCEQ domain scores.

The following analyses will be conducted in only Group-2 PK analysis set:

• To test if the time to the maximum nicotine concentration in THS 2.2 is shorter than in NRT gum the following hypothesis will be evaluated:

D--- 05 - C120


$$H_0$$
:  $X_{THS}$  -  $X_{NRT}$ = 0  $H_A$ :  $X_{THS}$  -  $X_{NRT}$ < 0

where  $X_{THS}$  and  $X_{NRT}$  are the median values of the THS 2.2 and NRT gum, respectively. The  $t_{max}$  will be analyzed on the original scale using the Wilcoxon Signed-Rank Test with a type I error  $\alpha = 0.025$  (one-sided test), as values are ordinal/discrete, and the assumption of normality may be questionable.

• To determine if the rate and the amount of nicotine absorbed of the THS 2.2 is higher relative to NRT gum the following hypothesis will be tested for both C<sub>max</sub> and AUC<sub>(0-last)</sub> parameters:

$$H_0: X_{THS}/X_{NRT} = 1.0$$
  $H_A: X_{THS}/X_{NRT} > 1.0$ 

where  $X_{THS}$  and  $X_{NRT}$  are the adjusted geometrical means of THS 2.2 and NRT gum, respectively.  $H_0$  is rejected with a type I error  $\alpha = 0.025$  (one-sided test), if the lower bound of the 95% CI for the  $X_{THS}/X_{NRT}$  ratio is higher than 1.0.

# 12.6.4 Confirmatory Analyses

Not applicable.

# 12.6.5 Safety Endpoints

In general, all safety data will be listed and tabulated on the safety population by sequence, using the approach described in Section 12.1.3. Safety variables collected during exposure periods will also be reported by product exposure.

AE data will serve as the primary assessment of safety. Other safety variables monitored in this study include: respiratory symptoms (cough assessment, VAS, and Likert scales); vital signs (systolic and diastolic blood pressure, pulse rate, respiratory rate); spirometry; ECG data; clinical chemistry, hematology, and urine analysis safety panel; physical examination; and concomitant medications.

The number and percentage of subjects with AEs and SAEs will be tabulated by system organ class and preferred term. Summaries will also be presented for AEs leading to withdrawal, AEs leading to Death, AEs by relatedness to product exposure, AEs by severity, and laboratory AEs. Tabulations will be performed for both the number of subjects experiencing an event and the number of events. The number and percentage of device events and of subjects with device events will be tabulated by sequence.

The number and percentage of subjects with clinical findings will be tabulated by sequence for laboratory parameters. Shift tables showing change from baseline of clinical findings will be provided for: ECGs, physical examinations, and laboratory parameters (both shifts in

Clinical Study Protocol Final 1.0 / 21 June 2013 Confidential


normal ranges and toxicity grades). Descriptive statistics will be summarized by visit and change from baseline for laboratory parameters, ECG, respiratory symptoms, and vital signs.

# 12.7 Exploratory Analyses

There are no planned exploratory analyses.

# 12.8 Interim Analysis

There are no planned interim analyses.

### 13 ADMINISTRATIVE CONSIDERATIONS

# 13.1 Principal Investigators and Study Administrative Structure

## 13.1.1 Principal Investigator

| Principal Investigator: | Koganeibashi Sakura Clinic |
|---|---|
| Masayuki Sugimoto M.D., Ph.D. | 2-11-25, Sakuracho, Koganei-shi, Tokyo 184-0005<br>Japan |
| | TEL:+81-<br>FAX: +81 |

Clinical Study Protocol Final 1.0 / 21 June 2013 Confidential


# 13.1.2 Sponsor

| Sponsor: | Philip Morris Products S.A |
|-----------------------------|-----------------------------------|
| | Quai Jeanrenaud 5, 2000 Neuchâtel |
| | Switzerland. |
| | Phone: +41 (58) 242 2111 |
| | Fax: +41 (58) 242 2811 |
| , PhD | Phone: +41 |
| Manager Clinical Science | Mobile: +41 |
| | E-mail: @pmi.com |
| , PhD | Phone: +41 |
| Staff Scientist, Statistics | Mobile: +41 |
| | Email: @pmi.com |
| , MD | Phone: +41 |
| Medical Safety Officer | Mobile: +41 |
| | E-mail: @pmi.com |
| | Phone: +41 |
| Medical Writer | Mobile: +41 |
| | Email: @pmi.com |
| , MSc | Phone: +41 |
| Clinical Study Manager | Mobile: +41 |
| | E-mail: @pmi.com |

Clinical Study Protocol Final 1.0 / 21 June 2013 Confidential


### 13.1.3 Other Responsibilities



(b) (4) is the local Contract Research Organization designated by PMI to manage and monitor the study: all duties and responsibilities transferred to (b) (4) by PMI will be defined in the agreement signed between the two parties

```
(b) (4)
```

```
(b) (4)
```

Any SAEs or pregnancies will be handled by:



Details of the laboratories conducting the clinical safety laboratory services, and biopharmaceutical analyses are shown in Appendix 2.

# 13.2 Subject Confidentiality

All information obtained during the conduct of the study with respect to the subjects' state of health will be regarded as confidential. A statement to this effect will be written in the information provided to the subject. An agreement to disclose any such information will be


obtained from the subject in writing and signed by the subject, in compliance with all local and national data protection and privacy legislation.

The anonymity of subjects participating in this study will be maintained. Subjects will be identifiable by the Sponsor (or Sponsor's authorized representative) on eCRFs and other documents by their subject (or randomization) number/code, sex and date of birth, but **not** by name, initial, or any other details relating to identifiable person (e.g. address, health insurance ID card, medical chart number, etc.). The assignment of a subject number/code for subject identification will be based on the appropriate data protection rules.

Any documents that allow full identification of the subject (e.g. the subject's signed ICF) must be maintained in confidence by the Investigator. If any document relating to this study shows a subject's name or any other details relating to an identifiable person (e.g. address, health insurance ID card, medical chart number, etc.), the name or other identifiable details must be obscured before a copy of that document is supplied to the Sponsor or the Sponsor's authorized representative.

#### 13.3 Access to Source Documentation

Subjects will be informed that, during the course of the clinical study, the Sponsor, any authorized representatives of the Sponsor, IRB, or regulatory authorities may inspect their medical records to verify the information collected, and ensure that all personal information made available for inspection is handled in the strictest confidence and in accordance with national and local data protection and privacy legislation.

The Investigator/head of the investigational site and all study site staff involved with the study must permit direct access to source data/documents for study related monitoring, audits, IRB review, and regulatory inspection(s).

#### 13.4 Record Retention

All records of data, source data and source documents (original records or certified copies), in any form (including, but not limited to, written, electronic, magnetic, optical records and scans, X-rays, and ECGs) that describe or record the methods, conduct, and/or results of the study, the factors affecting the study, and the actions taken will be maintained by the Principal Investigator/head of investigational site for the study, as required by ICH GCP and any other applicable local or national regulations. For X-rays at least the radiologist's assessment is required as source documentation. If the actual image is available it can be stored on CD as well.

Essential study documents/records, which individually and collectively permit evaluation of the conduct of a study and the quality of the data produced, are described in Article 41 of Ministerial Ordinance on GCP (Ordinance of the Ministry of Health and Welfare No. 28 of Confidentiality statement: Data and information contained in this document are considered to constitute trade secrets and confidential commercial information, and the legal protections provided to such trade secrets and confidential information are hereby claimed under the provisions of applicable law. No part of this document may be publicly disclosed without the written consent of Philip Morris Products S.A.


March 27, 1997 (as last amended by the Ordinance of Ministry of Health, Labour and Welfare No. 161 of December 28, 2012)),. Essential documents must be retained by the Principal Investigator/head of investigational site for a minimum of:

- At least 15 years after completion or discontinuation of the study, or
- At least 2 years depending on, for example, the circumstances, or
- After formal discontinuation of clinical development of the IP.

These documents should be retained for a longer period, however, if required by the applicable regulatory requirements or by an agreement with the Sponsor.

Examples of essential records/documents include, but are not limited to:

- Signed informed consent documents for all subjects and Master ICF.
- Subject identification code list, Screening Log and Enrolment Log (if applicable).
- Record of all communications between the Principal Investigator and the IRB, composition of the IRB.
- Record of all communications/contact between the Investigator, Sponsor, and its authorized representatives.
- List of sub-Investigators and other appropriately qualified persons to whom the head of the investigational site has delegated significant study-related duties, together with their roles in the study.
- Investigator Logs.
- eCRFs, study specific questionnaires (and associated data/scoring), subject diaries.
- Adverse event reports and details of follow-up investigations, details of concomitant medication
- All other Source Documents (e.g., chest X-rays, ECGs, consultation reports, physical examination, laboratory records) or any electronically captured study source data.
- Clinical laboratory reports, laboratory normal ranges.
- Original medical/hospital records, if applicable (the medical files of study subjects must be retained in accordance with local legislation and in accordance with the maximum period of time permitted by the hospital or study site).
- Record of any body fluids or tissue samples collected and retained.
- Device Issue Log, IP Accountability Logs, dispensing records.
- Information regarding subjects' discontinuation and any follow-up.


It is the responsibility of the Sponsor to inform the Principal Investigator/head of investigational site as to when these documents no longer need to be retained.

The Principal Investigator/head of investigational site must take measures to prevent accidental or premature destruction of these documents.

If the head of the investigational site wishes to assign the study records to another party or move them to another location, the Sponsor must be notified in advance.

The head of the investigational site must obtain written approval from the Sponsor before destruction of any records. Normally, these records will be held in the Investigator's archives. If the head of the investigational site is unable to meet this obligation, they must ask the Sponsor for permission to make alternative arrangements. Details of these arrangements must be documented.

The Sponsor's authorized representative will maintain documentation relating to the study as long as the IP is on the market, and/or for 15 years after the CSR has been finalized.

# 13.5 Clinical Study Report

The Sponsor must ensure that a CSR for this study is prepared regardless of whether the study is completed or prematurely terminated.

The CSR will be written based on standards of the ICH Guideline for the Structure and Content of Clinical Study Reports. In certain circumstances, an abbreviated CSR may be acceptable. Submission of the CSR to the IRB will be complied with as requested by local requirements.

The results of the additional variables for analysis will be presented in reports separate from the study CSR.

#### 13.6 Financial Disclosure

Investigators are required to provide financial disclosure information to the Sponsor. In addition, the Investigators must provide to the Sponsor a commitment to promptly update this information if any relevant changes occur during the course of the investigation and for 1 year following the completion of the study.

# 13.7 Publication and Disclosure Policy

This document contains data, information, and trades secretes that are confidential and proprietary to the Sponsor. This document is being provided solely for the purpose of

Clinical Study Protocol Final 1.0 / 21 June 2013 Confidential


evaluation and/or conducting this clinical study for the Sponsor. Disclosure of the content of this document is allowed only to study personnel, IRB, or duly authorized representatives of regulatory agencies for this purpose under the condition that confidentiality is maintained. The contents of this document may not be used in any other clinical study, disclosed to any other person or entity without the prior written permission of the Sponsor. The foregoing shall not apply to disclosure required by any regulations; however, prompt notice will be given to the Sponsor prior to any such disclosure.

The Sponsor plans to disclose details of the study protocol on a web-based, publicly available, clinical trial register database (e.g., ClinicalTrials.gov).

### 13.8 Insurance

The Sponsor is responsible for AEs and health damage of the subjects that are associated with the THS 2.2 product or with study procedures which are used during the study, except for AEs and health damage of the subjects caused by a negligent or an intentional misconduct and/or significant deviation to the protocol of the Investigator or the clinical trial site or the subjects. The Sponsor has taken out insurance to cover any bodily injury and property damage caused by the operations cried out by the insured.


### 14 REFERENCE LIST

#### Beal, 1989

Beal SL. Sample Size Determination for Confidence Intervals on the Population Means and on the Difference between Two Population Means. 1989; Biometrics, 45, 969–977.

### Benowitz et al., 2002

SNRT subcommittee on biochemical verification. Biochemical verification of tobacco use and cessation. Nicotine Tob Res. 2002; 4 (2): 149-159.

### Benowitz et al., 2006

Benowitz NL, Lessov-Schlaggar CN, Swan GE, Jacob P 3rd. Female sex and oral contraceptive use accelerate nicotine metabolism. Clin Pharmacol Ther. 2006;79(5):480-488.

### Benowitz et al., 2009

Benowitz NL, Hukkanen J, Jacob P. Nicotine chemistry, metabolism, kinetics and biomarkers. Handb Exp Pharmacol. 2009;192:29-60.

#### Cappelleri et al., 2007

Cappelleri JC, Bushmakin AG, Baker CL, Merikle E, Olufade AO, Gilbert DG. Confirmatory factor analyses and reliability of the modified cigarette evaluation questionnaire. Addict Behav. 2007 May; 32 (5): 912-23.

### Cox et al., 2001

Cox LS, Tiffany ST, Christen AG. Evaluation of the brief questionnaire of smoking urges (QSU-brief) in laboratory and clinical settings. Nicotine Tob Res. 2001; 3 (1): 7-16.

#### Dautzenberg et al., 2007

Bertrand Dautzenberg, Mitchell Nides, Jean-Luc Kienzler and Anne Callens. Pharmacokinetics, safety and efficacy from randomized controlled trials of 1 and 2 mg nicotine bitartrate lozenges (Nicotinell®). BMC Clinical Pharmacology 2007, 7:11 doi:10.1186/1472-6904-7-11. Available at http://www.biomedcentral.com/content/pdf/1472-6904-7-11.pdf (accessed on 01 February 2013)

Philip Morris Products S.A.

ZRHR-PK-02-JP

Clinical Study Protocol Final 1.0 / 21 June 2013


Declaration of Helsinki, 2008

Declaration of Helsinki. World Medical Association. Available from: http://www.wma.net/en/30publications/10policies/b3/index.html (accessed on 21 March 2012).

### EMA, 2008

European Medicines Agency, Committee for Medicinal Products for Human Use (CHMP). Guideline on the investigation of bioequivalence. 2008. CHMP/EWP/QWP/1401/98 Rev. 1. Available at http://www.ema.europa.eu/docs/en\_GB/document\_library/Scientific\_guideline/-2009/09/WC500003011.pdf

### Fagerström et al., 2012

Fagerström K, Russ C, Yu C, Yunis C and Foulds J. The Fagerström Test for Nicotine Dependence as a Predictor of Smoking Abstinence: A Pooled Analysis of Varenicline Clinical Trial. Nicotine & Tobacco Research. 2012; first published online March 30, 2012.

### Fagerström and Schneider, 1989

Fagerström KO, Schneider NG. Measuring nicotine dependence: a review of the Fagerström Tolerance Questionnaire. Journal of Behavioral Medicine. 1989; 12: 159-181.

#### FDA, 2001

United States Food and Drug Administration, Center for Drug Evaluation and Research. Statistical Approaches to Establishing Bioequivalence. January 2001.

Available from http://www.fda.gov/downloads/Drugs/.../Guidances/ucm070244.pdf

#### FDA, 2002

United States Food and Drug Administration. Guidance for Industry, Food-Effect Bioavailability and Fed Bioequivalence Studies, 2002. Available from http://www.fda.gov/cder/guidance/index.htm (accessed on 26 Sep 2012).

## FDA, 2011

United States Food and Drug Administration, Harmful and Potentially Harmful Constituents in Tobacco Products and Tobacco Smoke; Request for Comments (76 FR 50226, Aug. 12, 2011).

Philip Morris Products S.A.

Clinical Study Protocol Final 1.0 / 21 June 2013


#### FDA, 2012a

ZRHR-PK-02-JP

United States Food and Drug Administration, Center for Tobacco Products. Modified Risk Tobacco Product Applications: Draft Guidance for Industry, March 2012. Available from <a href="http://www.fda.gov/TobaccoProducts/GuidanceComplianceRegulatoryInformation/default.htm">http://www.fda.gov/TobaccoProducts/GuidanceComplianceRegulatoryInformation/default.htm</a>.

### FDA, 2012b

United States Food and Drug Administration. Implementation Specifications, reporting medical device problems, C54451/Medical Device Problem Codes, FDA, CDRH. Available from http://www.fda.gov/MedicalDevices/Safety/ReportaProblem/EventProblemCodes/ucm135741.htm# (accessed on 04 October 2012).

#### FDA, 2012c

United States Food and Drug Administration, Center for Tobacco Products. Modified Risk Tobacco Product Applications: Draft Guidance for Industry, March 2012. Fleiss et al, 1985

Fleiss JL, Wallenstein S, Rosenfeld R. Adjusting for baseline measurements in the two-period crossover study: a cautionary note. Control Clin Trials. 1985 Sep;6(3):192-7.

### Hatsukami et al., 2007

D.K. Hatsukami, A.M. Joseph, M. Lesage, J. Jensen, S.E. Murphy, P.R. Pentel, M. Kotlyar, E. Borgida, C. Le, and S.S. Hecht, Developing the science base for reducing tobacco harm, 9(4) Nicotine & Tobacco research S537 (Dec. 2007).

#### Health Canada, 1999

Health Canada. Determination of "Tar", Nicotine and Carbon, Monoxide in Mainstream Tobacco Smoke. Available at www.hc-sc.gc.ca.

#### Honjo et al., 2010a

Honjo K, Iso H, Tsugane S, Tamakoshi A, Satoh H, Tajima K et al. The effects of smoking and smoking cessation on mortality from cardiovascular disease among Japanese: pooled analysis of three large-scale cohort studies in Japan. Tob Control. 2010; 19 (1): 50-57.

#### Honjo et al., 2010b

Honjo K, Iso H, Inoue M, Tsugane S; JPHC Study Group. Smoking cessation: predictive factors among middle-aged Japanese. Nicotine Tob Res. 2010; 12 (10): 1050-1054.

Clinical Study Protocol Final 1.0 / 21 June 2013


#### ICH E9, 1998

European Medicines Agency. ICH Topic E9: Statistical Principles for Clinical Trials (CPMP/ICH/363/96 – adopted March 1998). Available at http://www.fda.gov/downloads/-Drugs/GuidanceComplianceRegulatoryInformation/Guidances/ucm073137.pdf.

### **Institute of Medicine, 2012**

Institute of Medicine Consensus Report. Scientific Standards for Studies on Modified Risk Tobacco Products. Released: December 14, 2011.Board on Population Health and Public Health Practice. (http://www.iom.edu/Reports/2011/Scientific-Standards-for-Studies-on-Modified-Risk-Tobacco-Products.aspx).

### **International Tobacco Online, 2012**

http://www.internationaltobaccoonline.com/japanese-survey-said-the-percentage-of-smokers-in-japan-is-lower-than-20-p-927.html (accessed 19 June 2012).

### Iso et al., 2005

Iso H, Date C, Yamamoto A, Toyoshima H, Watanabe Y, Kikuchi S et al.; JACC Study Group. Smoking cessation and mortality from cardiovascular disease among Japanese men and women: the JACC Study. Am J Epidemiol. 2005; 161 (2): 170-179.

#### Jacob et al., 2011

Jacob P 3rd, Yu L, Duan M, Ramos L, Yturralde O, Benowitz NL. Determination of the Nicotine Metabolites Cotinine and *Trans-3'-Hydroxycotinine* in Biologic fluids of Smokers and Non-smokers using Liquid Chromatography - Tandem Mass Spectrometry: Biomarkers for Tobacco Smoke Exposure and for Phenotyping Cytochrome P450 2A6 Activity. J Chromatogr B Analyt Technol Biomed Life Sci. 2011 Feb 1; 879 (3-4): 267-76.

#### Lacy et al., 2007

Lacy CF, Armstrong LL, Goldman MP, Lance LL eds. Drug Information Handbook 15th ed. Hudson, OH; LexiComp Inc. 2007: 1899-1912.

#### Lingling, 2008

Lingling Han, Merck & Co., Inc., North Wales, PA. Calculating the point estimate and confidence interval of Hodges-Lehmann's median using SAS® software. Paper ST-154, SESUG Proceedings. Available from http:// analytics.ncsu.edu/sesug/2008/ST-154.pdf (accessed on 04 Oct 2012)

Clinical Study Protocol Final 1.0 / 21 June 2013


#### Matta et al., 2006

Matta SG, Balfour DJ, Benowitz NL, Boyd RT, Buccafusco JJ, Caggiula AR et al. Guidelines on nicotine dose selection for in vivo research. Psychopharmacology (Berl). 2007; 190 (3): 269-319.

### Ministry of Health, Labour and Welfare, 1997

Ministerial Ordinance on Good Clinical Practice for Drugs, Ordinance of the Ministry of Health and Welfare No. 28 of March 27, 1997, as last amended by the Ordinance of Ministry of Health, Labour and Welfare No. 161 of December 28, 2012.

#### PMI, 2012

Philip Morris International, 2012. In French. Work Instruction PMI\_RD\_WKI\_000527: Guide d'utilisation de l'extracteur in situ, nettoyage des seringues, des pistons, des aiguilles et des pieges (R2540.M109). Version 3.0.

### PMI, 2013a

Philip Morris International. 2013. Internally-modified method based on International Organization for standardization's ISO 4387:2000. In French. PMI\_RD\_WKI\_000530: Détermination du TMP et CO et trappage de l'eau, nicotine, acide pyruvique et des smoke constituents:BaP, phénols, TSNA et amines aromatiques.

### PMI, 2013b

Philip Morris International, Neuchatel, Switzerland, 2013. Investigator's Brochure for Tobacco Heating System 2.2.

### PMI, 2013c

Philip Morris International. 2013. David Ghosh. Experimental report: Identifying the appropriate technique to collect and extract water, nicotine and glycerin from the TPM to further characterize the tar of the ZURICH product. Version 1.0.

# **PMI White Paper Docket**

Food and Drug Administration (FDA), Division of Dockets Management. Philip Morris's International comments on the scientific evaluation of the modified risk tobacco product applications. Docket no. FDA-2011-N-0443.

Clinical Study Protocol Final 1.0 / 21 June 2013


### Rodgman and Perfetti, 2009

A. Rodgman, and T.A. Perfetti, the chemical components of tobacco and tobacco smoke (Taylor & Francis Group 2009).

## Senn, 2002

Senn S. Cross-over Trials in Clinical Research. 2002; John Wiley & Sons. ISBN: 978-0-471-49653-3

### Shiffman et al., 2004

Shiffman S, West R, Gilbert D; SRNT Work Group on the Assessment of Craving and Withdrawal in Clinical Trials. Recommendation for the assessment of tobacco craving and withdrawal in smoking cessation trials. Nicotine Tob Res. 2004 Aug;6(4):599-614.

## Tiffany et al., 1991

Tiffany ST, Drobes DJ. The development and initial validation of a questionnaire on smoking urges. British Journal of Addiction. 1991; 86: 1467-1476.

#### WHO, 2002

Evidence Based Recommendations on the Treatment of Tobacco Dependence. June 2001.

### Zeller and Hatsukami, 2009

Zeller M, Hatsukami D; Strategic Dialogue on Tobacco Harm Reduction Group. The Strategic Dialogue on Tobacco Harm Reduction: a vision and blueprint for action in the US. Tob Control. 2009; 18.

#### ZRHX-PK-02, 2012

Philip Morris International, Switzerland. 2012. Clinical study. A Single-center, Open-label, Randomized, Controlled, Crossover Study to Explore the Nicotine Pharmacokinetic Profile and Safety of Tobacco Heating System (THS) 2.1 Compared to Conventional Cigarettes Following Single and ad Libitum Use in Smoking, But Otherwise Healthy Subjects. Available at http://clinicaltrials.gov/ct2/show/NCT01780688?term=NCT01780688&rank=1
Clinical Study Protocol Final 1.0 / 21 June 2013


# Appendix 1 Schedule of Events

| | Screening | Admission | Wash-<br>out | Single<br>use | Wash-out | Single<br>use | Day of<br>Discharge <sup>k</sup> | Safety follow-up |
|---|---|---|---|---|---|---|---|---|
| Study Day | -29 to -2 | -1 | 0 | 1 | 2 | 3 | 4 | 4 to 11 |
| Informed consent/subject information sheet | • | | | | | | | |
| Advice on the risks of smoking and debriefing | • | • | | | | | • | |
| Inclusion/exclusion criteria | • | • | | | | | | |
| Enrolment | | • | | | | | | |
| Randomization | | | • | | | | | |
| Product demonstration of THS 2.2 and NRT gum | • | | | | | | | |
| Product test for THS 2.2 and NRT gum | | • | | | | | | |
| Product use | | | | • | | • | | |
| Support during periods of reduced smoking/smoking abstinence (as required) | | | • | • | • | • | | |
| Identification of current CC brand | • | • | | | | | | |
| Smoking history | • | • | | | | | | |

Clinical Study Protocol Final 1.0 / 21 June 2013


| | Screening | Admission | Wash-<br>out | Single<br>use | Wash-out | Single<br>use | Day of<br>Discharge <sup>k</sup> | Safety follow-up |
|---|---|---|---|---|---|---|---|---|
| Study Day | -29 to -2 | -1 | 0 | 1 | 2 | 3 | 4 | 4 to 11 |
| Readiness to abstain from smoking for up to 4 days | • | • | | | | | | |
| Willingness to quit smoking in the next 3 months | • | | | | | | | |
| Demographics <sup>a</sup> , medical history, concomitant diseases | • | | | | | | | |
| Prior medication <sup>b</sup> / Concomitant medication | • | • | • | • | • | • | • | • |
| Physical examination, body<br>height, weight and related BMI <sup>c</sup> | • | • | | | | | • | |
| Vital signs <sup>d</sup> | • | • | • | • | • | • | • | |
| ECG | • | | | • | | • | | |
| Spirometry | • | • | | | | | • | |
| Chest X-ray <sup>e</sup> | • | | | | | | | |
| B/U: Hematology, clinical chemistry, urine analysis | • | • | | | | | • | |
| B: Serology | • | | | | | | | |
| U: Urine drug screen, urine cotinine screen | • | • | | | | | | |
| Alcohol test | • | • | | | | | | |
| U: Pregnancy test (all females) | • | • | | | | | • | |

Clinical Study Protocol Final 1.0 / 21 June 2013


| | Screening | Admission | Wash-<br>out | Single<br>use | Wash-out | Single<br>use | Day of<br>Discharge <sup>k</sup> | Safety follow-up |
|---|---|---|---|---|---|---|---|---|
| Study Day | -29 to -2 | -1 | 0 | 1 | 2 | 3 | 4 | 4 to 11 |
| Collection of used Tobacco<br>Sticks and CC butts and NRT<br>gum | | | | • | | • | | |
| B: Plasma nicotine <sup>f</sup> | | | | • | • | • | • | |
| B: COHb <sup>g</sup> | | | | • | | • | | |
| B. 00110 | | | | (5x) | | (5x) | | |
| CO breath test h | | • | • | • | • | • | • | |
| | | (1x) | (4x) | (4x) | (4x) | (4x) | (1x) | |
| B: trans-3'-hydroxycotinine and cotinine (CYP2A6 activity) in plasma | | • | | | | | | |
| FTND questionnaire | • | | | | | | | |
| QSU-brief questionnaire i | | | | • | | • | | |
| MCEQ (modified version, only after THS 2.2 and CC use | | | | • | | • | | |
| Cough assessment j | | | • | • | • | • | • | |
| AE/SAE recording | • | • | • | • | • | • | • | • |

Abbreviations: AE = Adverse event; BMI = Body mass index; CC = Conventional cigarette(s); CO = Carbon monoxide; COHb = Carboxyhemoglobin; CYP2A6 = Cytochrome P450 2A6; ECG = Electrocardiogram; FTND = Fagerström Test for Nicotine Dependence (revised version); MCEQ = Modified Cigarette Evaluation Questionnaire; NRT gum = Nicotine replacement therapy gum; QSU-brief = Questionnaire of Smoking Urges brief; SAE = Serious adverse event; THS 2.2 = Tobacco Heating System 2.2

B: Blood sample required.

U: Urine sample required.

#### a: Sex, date of birth/age.

Philip Morris Products S.A.

Clinical Study Protocol


ZRHR-PK-02-JP

Final 1.0 / 21 June 2013


- b: Prior medication at Screening and the 4 weeks prior to Screening.
- c: Including height (only at Screening), body weight and calculated BMI.
- d: Systolic and diastolic blood pressure, pulse rate, respiratory rate.
- e: Pre-study chest X-ray (anterior-posterior and left lateral views) to be used, if performed within 6 months prior to Screening.
- f: Nicotine blood samples to be taken as follows:

#### Single Use on Day 1 and Day 3 for THS 2.2 and CC only:

For subjects on THS 2.2 or on CC, a total of 16 blood samples will be taken for a 24-hour profile (Day 1 and Day 3). The first blood sample will be taken within 15 minutes prior to the single use ( $T_0$ ). Times of sampling are thereafter in relation to  $T_0$ :  $T_1$  after 2 minutes + 1 min,  $T_2$  after 4 minutes + 1 min,  $T_3$  after 6 minutes + 1 min,  $T_4$  after 8 minutes + 1 min,  $T_5$  after 10 minutes + 1 min,  $T_6$  after 15 minutes + 2 min,  $T_7$  after 30 minutes + 2 min,  $T_8$  after 45 minutes + 2 min,  $T_9$  after 60 minutes + 3 min,  $T_{10}$  after 2 hours + 5 min,  $T_{11}$  after 12 hours + 5 min,  $T_{12}$  after 6 hours + 5 min,  $T_{13}$  after 9 hours + 5 min,  $T_{14}$  after 12 hours + 5 min, and  $T_{15}$  after 24 hours + 5 min (this sample will be drawn during the day following product use, i.e., wash-out).

#### Single Use on Day 1 and Day 3 for NRT gum only:

For subjects on NRT gum: A total of 16 blood samples will be taken for a 24-hour profile (Day 1 and Day 3). The first blood sample will be taken within 15 min  $T_0$ , Thereafter in relation to  $T_0$ :  $T_1$  after 10 min + 1 min,  $T_2$  after 20 minutes + 1 min,  $T_3$  after 25 minutes + 1 min,  $T_4$  after 30 minutes + 1 min,  $T_5$  after 35 minutes + 1 min,  $T_6$  after 40 minutes + 1 min,  $T_7$  after 45 minutes + 1 min,  $T_8$  after 60 minutes + 3 min,  $T_9$  after 2 hours + 5 min,  $T_{10}$  after 3 hours + 5 min,  $T_{11}$  after 4 hours + 5 min,  $T_{12}$  after 6 hours + 5 min,  $T_{13}$  after 9 hours + 5 min,  $T_{14}$  after 12 hours + 5 min, and  $T_{15}$  after 24 hours + 5 min (this sample will be drawn during the day following product use, i.e., wash-out).

#### g: COHb blood samples to be taken as follows:

Single use: A total of 5 blood samples will be taken. The first sample within 15 minutes prior to T0 (start of single product use); thereafter in relation to T0 at 15 min +2 min, 60 min +3 min, 4 hours +5 min and 12 hours +5 min.

- h: A CO breath test will be conducted once on Day -1 and Day 4. On Day 0, Day 1, Day 2, Day 3, four breath tests will be done per day. On Day 1 and Day 3, the first test per day will be performed within 15 minutes prior to T<sub>0</sub> (T<sub>0</sub> = start of first product use) the three other tests will be conducted as described in section 9. On the wash-out days (Day 0 and Day 2) the first test will be conducted between 8:00 am-09:30 am, the three other test will be conducted as described as section 9.
- i: QSU-brief will be assessed as follows:

Single use: The QSU-brief will be completed by the subject himself/herself at single use study days.

THS 2.2 and CC arms: First sample within 15 min prior to T<sub>0</sub>, 9 assessments thereafter in relation to T<sub>0</sub>: 15 min, 30 min, 45 min, 60 min, 2 hr, 4 hrs, 6 hrs, 9 hrs, and 12 hrs after T<sub>0</sub> with a time window of 10 minutes each.

NRT arm: First sample within 15 min prior to T<sub>0</sub>, 9 assessments thereafter in relation to T<sub>0</sub>: 20 min, 30 min, 45 min, 60 min, 2 hr, 4 hr, 6 hrs, 9 hrs, and 12 hrs after T<sub>0</sub> with a time window of 10 minutes.

- j: Visual analogue scale, three Likert scales and one open question.
- k: All examinations listed at the Day of Discharge should also be conducted in subjects preliminarily terminating the study.
- I: Spontaneous reporting of new AEs/SAEs by the subject and active follow-up of ongoing AEs/SAEs by the site.

Clinical Study Protocol Final 1.0 / 21 June 2013 Confidential


# **Appendix 2** Participating Laboratories

The following Laboratories will be used in the study:

## **CELERION (USA and Switzerland)**

USA: Celerion, 621 Rose Street, 68502, Lincoln, NE, USA

Switzerland: Celerion, Allmendstrasse 32, 8320 Fehraltorf, Switzerland



## TOKIWA CHEMICAL INDUSTRIES CO.,LTD.

16-22, Kamiikebukuro 4-chome, Toshima-ku, Tokyo, 170-0012, Japan

More details will be found in the study laboratory manuals.

Clinical Study Protocol Final 1.0 / 21 June 2013 Confidential


# **Appendix 3** Investigational Product and Instructions for Use

The product user guide will be provided as a separate document.

Clinical Study Protocol Final 1.0 / 21 June 2013 Confidential


# Appendix 4 THS Package Label

The package label for the THS Tobacco Sticks (example):



Clinical Study Protocol Final 1.0 / 21 June 2013 Confidential


Clinical Study Protocol Final 1.0 / 21 June 2013


The package label for the THS Tobacco Sticks carton (example):




# Appendix 5 Abnormal Laboratory Values

# ABNORMAL LABORATORY VALUES RATING: SERUM CHEMISTRY PARAMETERS

| Serum Chemistry* | Mild | Moderate | Severe |
|---|---|---|---|
| | (Grade 1) | (Grade 2) | (Grade 3) |
| Sodium – Hyponatremia (mmol/l) ** (1) | <lln -="" 130<="" td=""><td>-</td><td>&lt;130 - 120</td></lln> | - | <130 - 120 |
| Sodium – Hypernatremia (mmol/l) ** (1) | >ULN - 150 | >150 - 155 | >155 - 160;<br>hospitalization<br>indicated |
| Potassium – Hyperkalaemia (mmol/l)** <sup>(1)</sup> | >ULN - 5.5 | >5.5 - 6.0 | >6.0 - 7.0;<br>hospitalization<br>indicated |
| Potassium – Hypokalaemia (mmol/l) ** <sup>(1)</sup> | <lln -="" 3.0<="" td=""><td><lln -="" 3.0;<br="">symptomatic;<br/>intervention indicated</lln></td><td>&lt;3.0 - 2.5;<br/>hospitalization<br/>indicated</td></lln> | <lln -="" 3.0;<br="">symptomatic;<br/>intervention indicated</lln> | <3.0 - 2.5;<br>hospitalization<br>indicated |
| Glucose – Hypoglycaemia ** <sup>(1)</sup> (mg/dL) | <lln 55;<="" td="" –=""><td>&lt;55 – 40;</td><td>&lt;40 – 30;</td></lln> | <55 – 40; | <40 – 30; |
| (mmol/l) | <lln 3.0<="" td="" –=""><td>&lt;3.0 – 2.2</td><td>&lt;2.2 – 1.7</td></lln> | <3.0 – 2.2 | <2.2 – 1.7 |
| Blood Urea Nitrogen (BUN) (mg/dL) (2) | 23 – 26 | 27 – 31 | >31 |
| Glucose – Hyperglycaemia: ** | | | |
| | >ULN – 160; | >160 -250 | >250 – 500; |
| Fasting <sup>(1)</sup> ((mg/dL) | >ULN - 8.9 | > 8.9-13.9 | >13.9 – 27.8 |
| (mmol/l) | | | Hospitalization indicated |
| Creatinine increased** (1) | >1 – 1.5 x baseline; | >1.5 – 3.0 x baseline; | >3.0 x baseline; |
| | >ULN – 1.5 x ULN | >1.5 – 3.0 x ULN | >3.0 – 6.0 x ULN |
| Albumin – Hypoalbuminaemia** <sup>(1)</sup> (g/dL) | <lln 3;<="" td="" –=""><td>&lt;3 – 2;</td><td>&lt;2;</td></lln> | <3 – 2; | <2; |
| (g/l) | <lln -="" 30<="" td=""><td>&lt;30 - 20</td><td>&lt;20</td></lln> | <30 - 20 | <20 |
| Total Protein – Hypoproteinaemia (2) | | | |
| (g/dL) | 5.5 – 6.0 | 5.0 – 5.4 | <5.0 |
| Alkaline phosphatase increased** (1) | >ULN – 2.5 x ULN | >2.5 – 5.0 x ULN | >5.0 – 20.0 x ULN |
| ALT / AST increased** (1) | >ULN – 3.0 x ULN | >3.0 – 5.0 x ULN | >5.0 – 20.0 x ULN |
| Gamma-glutamyl transferase | >ULN – 2.5 x ULN | >2.5 – 5.0 x ULN | >5.0 – 20.0 x ULN |
| increased <sup>(1)</sup> | | | |

Clinical Study Protocol Final 1.0 / 21 June 2013


| Blood bilirubin increased ** (1) | >ULN – 1.5 x ULN | >1.5 – 3.0 x ULN | >3.0 – 10.0 ULN |
|---|---|---|---|
| Cholesterol high** (1) (mg/dL) (mmol/l) | >ULN – 300; | >300-400; | >400-500; |
| | >ULN – 7.75 | >7.75-10.34 | >10.34-12.92 |
| Triglycerides - Hypertriglyceridemia <sup>(1)</sup> (mg/dL) (mmol/l) | 150 – 300; | >300 – 500; | >500 – 1000; |
| | 1.71 – 3.42 | >3.42 – 5.70 | >5.70 – 11.40 |

Abbreviations: ALT = Alanine aminotransferase; AST = Aspartate aminotransferase; LLN = Lower limit of the normal range; ULN = Upper limit of the normal range.

#### Data Sources:

- (1) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, U.S. Department of Health and Human Services, Food and Drug Administration (FDA), Center for Biologics Evaluation and Research Guidance for Industry.
- (2) Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, U.S. Department of Health and Human Services, FDA, Center for Biologics Evaluation and Research Guidance for Industry.
- \* Those parameters that are not listed do not have grading categories in either the CTCAE or the FDA guidance documents and will therefore be reviewed by the Investigator and only reported as an AE if considered to be clinically relevant.
- \*\* Where parameters in this table are listed in both the CTCAE and the FDA guidance documents, and each document has different values within each grading category, the grading in CTCAE guidance document predominates.

ZRHR-PK-02-JP

Final 1.0 / 21 June 2013

### ABNORMAL LABORATORY VALUES RATING: HEMATOLOGY PARAMETERS

| Haematology* | Mild | Moderate | Severe |
|---|---|---|---|
| | (Grade 1) | (Grade 2) | (Grade 3) |
| Haemoglobin (Female) – (g/dL) (1) | 11.0 – 12.0 | 9.5 – 10.9 | 8.0 – 9.4 |
| change from baseline value – (g/dL) <sup>(1)</sup> | Any decrease – 1.5 | 1.6 – 2.0 | 2.1 – 5.0 |
| Haemoglobin (Male) – (g/dL) <sup>(1)</sup> | 12.5 – 13.5 | 10.5 – 12.4 | 8.5 – 10.4 |
| change from baseline value – (g/dL) <sup>(1)</sup> | Any decrease – 1.5 | 1.6 – 2.0 | 2.1 – 5.0 |
| Haemoglobin increase – (g/dL) <sup>(2)</sup> | Increase in >0 – 2<br>above ULN or<br>above baseline if<br>baseline is above<br>ULN | Increase in >2 – 4<br>above ULN or<br>above baseline if<br>baseline is above<br>ULN | Increase in >4 above ULN or above baseline if baseline is above ULN |
| WBC Increase – (cell/mm <sup>3</sup> ) (1) | 10,800 – 15,000 | 15,001 – 20,000 | 20,001 – 25,000 |
| WBC Decrease - (cell/mm <sup>3</sup> ) (2)** | <lln 3000;<="" td="" –=""><td>&lt;3000 - 2000;</td><td>&lt;2000 - 1000;</td></lln> | <3000 - 2000; | <2000 - 1000; |
| | <lln -="" 10<sup="" 3.0="" x="">-9/l</lln> | <3.0 – 2.0 x 10 <sup>-9</sup> /l | <2.0 – 1.0 x 10 <sup>-9</sup> /l |
| Lymphocytes Increase - (cell/mm <sup>3</sup> ) (2) | - | >4,000 – 20,000 | >20,000 |
| Lymphocytes Decrease - (cell/mm³) (2)** | <lln 800;<="" td="" –=""><td>&lt;800 - 500;</td><td>&lt;500 - 200;</td></lln> | <800 - 500; | <500 - 200; |
| | <lln 0.8="" 10<sup="" x="" –="">-9/l</lln> | <0.8 – 0.5 x 10 <sup>-9</sup> /l | <0.5 – 0.2 x 10 <sup>-9</sup> /l |
| Neutrophils Decrease - (cell/mm³) (2)** | <lln 1500;<="" td="" –=""><td>&lt;1500 - 1000;</td><td>&lt;1000 - 500;</td></lln> | <1500 - 1000; | <1000 - 500; |
| | <lln 1.5="" 10<sup="" x="" –="">-9/l</lln> | <1.5 – 1.0 x 10 <sup>-9</sup> /l | <1.0 – 0.5 x 10 <sup>-9</sup> /l |
| Eosinophils - (cell/mm <sup>3</sup> ) (1) | 650 – 1500 | 1501 - 5000 | >5000 |
| Platelets Decrease - (cell/mm³) (2)** | <lln 75,000;<="" td="" –=""><td>&lt;75,000 – 50,000;</td><td>&lt;50,000 – 25,000;</td></lln> | <75,000 – 50,000; | <50,000 – 25,000; |
| | <lln 10<sup="" 75.0="" x="" –="">-9/l</lln> | <75.0 – 50.0 x 10 <sup>-9</sup> /l | <50.0 – 25.0 x 10 <sup>-9</sup> /l |

Abbreviations: LLN = Lower limit of the normal range; ULN = Upper limit of the normal range; WBC = White blood cell (count).

Data Source: (1) Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, U.S. Department of Health and Human Services, FDA, Center for Biologics Evaluation and Research - Guidance for Industry.

(2) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.

Clinical Study Protocol Final 1.0 / 21 June 2013


\* Those parameters that are not listed do not have grading categories in either the CTCAE or the FDA guidance documents and will therefore be reviewed by the Investigator and only reported as an AE if considered to be clinically relevant.

\*\* Where parameters in this table are listed in both the CTCAE and the FDA guidance documents, and each document has different values within each grading category, the grading in CTCAE guidance document predominates.

Clinical Study Protocol Final 1.0 / 21 June 2013 Confidential


#### ABNORMAL LABORATORY VALUES RATING: URINALYSIS PARAMETERS

| Urine* | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) |
|---|---|---|---|
| Protein ** (1) | 1+ proteinuria;<br>urinary protein<br><1.0 g/24 hours | 2+ proteinuria;<br>urinary protein<br>1.0-3.4 g/24 hours | Urinary protein<br>≥3.5 g/24 hours |
| Glucose (2) | Trace | 1+ | 2+ |
| Blood – Haematuria ** <sup>(1)</sup> | Asymptomatic;<br>clinical or<br>diagnostic<br>observations<br>only;<br>intervention not<br>indicated | Symptomatic;<br>urinary catheter or<br>bladder irrigation<br>indicated; limiting<br>instrumental ADL | Gross haematuria; transfusion, IV medications or hospitalization indicated; elective endoscopic, radiologic or operative intervention indicated; limiting self-care ADL |

Abbreviations: ADL = Activities of daily living; IV = Intravenous.

Data Source: (1) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.

- (2) Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, U.S. Department of Health and Human Services, FDA, Center for Biologics Evaluation and Research Guidance for Industry.
- \* Those parameters that are not listed do not have grading categories in either the CTCAE or the FDA guidance documents and will therefore be reviewed by the Investigator and only reported as an AE if considered to be clinically relevant.
- \*\* Where parameters in this table are listed in both the CTCAE and the FDA guidance documents, and each document has different values within each grading category, the grading in CTCAE guidance document predominates.



# ZRHR-PK-02-JP **Clinical Study Protocol** Signature Pages

Study Title:

A single-centre, open-label, randomized, controlled, crossover study to investigate the nicotine pharmacokinetic profile and safety of Tobacco Heating System 2.2 (THS 2.2) following single use in smoking, healthy subjects compared to

conventional cigarettes and nicotine gum

Study Number:

ZRHR-PK-02-JP

**Product Name:** 

Tobacco Heating System 2.2 (THS 2.2)

Principal Investigator and

Masayuki Sugimoto M.D., Ph.D.

Affiliation:

Koganeibashi Sakura Clinic

2-11-25, Sakuracho, Koganei-shi,

Tokyo 184-0005 Japan

Sponsor:

Philip Morris Products S.A.

Quai Jeanrenaud 5

2000 Neuchâtel

**Sponsor Signatories:** 

PhD, Manager Clinical Science

, PhD, Biostatistician

, MD, Medical Safety Officer

Version:

Final 1.0

Date:

21 June 2013

Confidentiality Statement

Philip Morris Products S.A.

Clinical Study Protocol


ZRHR-PK-02-JP

Version Final 1.0 / 21th of June

Page 2 of 3

## PRINCIPAL INVESTIGATOR'S SIGNATURE

### PRINCIPAL INVESTIGATOR'S SIGNATURE

Study Title:

A single-centre, open-label, randomized, controlled, crossover study to investigate the nicotine pharmacokinetic profile and safety of Tobacco Heating System 2.2 (THS 2.2) following single use in smoking, healthy subjects compared to conventional cigarettes and nicotine gum

Study Number:

ZRHR-PK-02-JP

I have read the protocol described above. I agree to comply with all applicable regulations and to conduct the study as described in the protocol.

By signing the protocol, the Investigator agrees to keep all information and documents provided by the Sponsor in strict confidence and to request similar confidentiality from his/her staff. The information provided by the Sponsor to the investigator may not be disclosed to others without direct written authorization from the Sponsor, except to the extent necessary to obtain informed consent from subjects who wish to participate in the study.

Signed: Masagula Pujimoto

Date: 01 / Jul /2013

DR MASAYUKI SUGIMOTO M.D., PH.D.

Philip Morris Products S.A.

Clinical Study Protocol


ZRHR-PK-02-JP

Version Final 1.0 / 21th of June

Page 3 of 3

## SIGNATURES OF SPONSORS RESPONSIBLE PERSONNEL

**SPONSOR SIGNATORIES** 

**Study Title:** 

A single-centre, open-label, randomized, controlled, crossover study to investigate the nicotine pharmacokinetic profile and safety of Tobacco Heating System 2.2 (THS 2.2) following single use in smoking, healthy subjects compared to conventional cigarettes and nicotine gum

Study Number:

ZRHR-PK-02-JP

This Clinical Study Protocol was subject to critical review and has been approved by the Sponsor. The following personnel contributed to writing and/or approving this protocol:

| Signed: | PhD, Manager Clinical Science | Date:_ | 21 June 2017. |
|---------|-------------------------------|--------|---------------|
| Signed: | , PhD, Biostatistician | Date:_ | 25 JUNE 2013 |
| Signed: | , MD, Medical Safety Officer | Date:_ | 25 June 2013 |

**Study Title:** 



# **NOTE TO FILE (11-AUG-2014)**

Clinical Study: ZRHR-PK-02-JP

A single-center, open-label, randomized, controlled, crossover study to investigate the nicotine pharmacokinetic

profile and safety of Tobacco Heating System 2.2

(THS 2.2) following single use in smoking, healthy subjects

compared to conventional cigarettes and nicotine gum

All sites **Investigational Site:** 

Philip Morris Products S.A., Research & Development **Sponsor:** 

Quai Jeanrenaud 5, 2000 Neuchâtel, Switzerland

**Author:** 

Updated Table 4 CYP2A6: Substrates, Inhibitors, and **Subject** 

Inducers

**Purpose** The purpose of this note to file is to inform that Table 4 "CYP2A6: Substrates, Inhibitors, and Inducers", which is a part of all Clinical Studies Protocols of P1 is updated in accordance with the Drug Information Handbook, 23d Edition.

**Background**: At the time of Clinical Protocols Development for P1, Table 4 created, with reference to the Drug Information Handbook 21d Edition. During Clinical Report preparation of the respective studies, the Table was revised based on the latest 23d Edition of 23d Edition of the Drug Information Handbook.

References Drug Information Handbook, 23d Edition

Table 4. CYP 2A6: Substrates, Inhibitors, Inducers

| Inhibitor | Drug Class |
|-----------------|-------------------------------|
| Amiodarone | Antiarrhythmic agent |
| Desipramine | Antidepressant |
| Isoniazid | Anti-bacterial drug |
| Ketoconazole | Anti-fungal agent |
| Letrozole | Anti-estrogen drug |
| Methoxsalen | Systemic psoralens |
| Miconazole | Anti-fungal agent |
| Tranylcypromine | Antidepressant |
| Inducer | Drug Class |
| Amobarbital | Barbiturates |
| Pentobarbital | Barbiturates |
| Phenobarbital | Barbiturates/anticonvulsant |
| Rifampin | Antimycobacterial |
| Secobarbital | Barbiturates |
| Substrate | Drug Class |
| Dexmedetomidine | α2-Adrenoceptor, sedative |
| Ifosfamide | Anti-cancer, alkylating agent |

| Name: Tamara Koval | Function Medical Safety Officer |
|--------------------|---------------------------------|

Signed: Date: 11 hugust 2014